#### STATISTICAL ANALYSIS PLAN

| Protocol No. | MT-1186-J01 |
|-----------------|--------------------------------------------------------|
| | Phase I Study of Oral Edaravone in Healthy Adult Males |
| Protocol Title | (Single- and Multiple-dose Study) |
| Version History | Version 1.0 First approved version / 7 September, 2018 |
| , <b>0.0.0</b> | Version 2.0 Final approved version / 9 October, 2018 |
| | <b>,</b> |

NCT number: NCT04481750

Author

#### APPROVAL FORM

The approval signatories below have reviewed this Statistical Analysis Plan (SAP) and agreed on the planned analyses defined in this document.

| ICRÓ Statistics / P | iai mācokinėtics Author(s). | |
|---|---|---|
| Name: | Date: | Signature: |
| Ivanic. | | |
| Position: | | |
| Responsible STA | Γ | |
| MTPC Statistics A | öprover | [MTPC-STATH] |
| Name: | Date: | Signature: |
| Position: | | |
| Head of regional | STAT | |
| MTPC Pharmacok | | [MTPC-STATH] |
| Name: | Date: | Signature: |
| Position: | | |
| Head of regional | on the end of the control of the property of the party of | and the second of the second o |
| MTPC Statistics R | eviewer ``\ | [MTPC-STATM] |
| Name: | Date: | Signature: |
| Position: | | |
| Responsible STA | T | AND THE RESERVE OF THE PROPERTY OF THE PROPERT |
| MTPC Pharmacok | | [MTPC-\$TATM] |
| Name: | Date: | Signature: |
| Position: | | |
| Responsible CP | | MTPC-STATI |
| MTPC Statistics R | eviewer<br>Ebiss | [WIFE-STAI] |
| Name: | Date: | Signature: |
| Position: | | |
| COT STAT | | |
| MTPC Pharmacol | ánetics Reviewer | [MTRG-STAT] |
| Name: | Date: | Signature: |
| Position: | | |
| COT CP | | |

#### TABLE OF CONTENTS

| 1. | INTI | TRODUCTION8 | |
|----|------|------------------------------------------------|----|
| | 1.1 | Study Design | 8 |
| | 1.2 | Schedule of Study Procedures | 8 |
| 2. | STU | DY OBJECTIVE(S) AND ENDPOINTS1 | 3 |
| | 2.1 | Study Objective(s) | 3 |
| | | 2.1.1 Primary Objective(s) | 3 |
| | | 2.1.2 Secondary Objectives | 3 |
| | 2.2 | Endpoints | 3 |
| | | 2.2.1 Safety Endpoints | .3 |
| | | 2.2.2 Pharmacokinetic Endpoints | .3 |
| | | 2.2.3 Pharmacodynamic Endpoints | .3 |
| 3. | PLA | NNED ANALYSES1 | 4 |
| 4. | ANA | ALYSIS POPULATION(S) <sup>1</sup> | 4 |
| 5. | GEN | NERAL CONSIDERATIONS | 4 |
| | 5.1 | .1 Subjects Composition14 | |
| | 5.2 | 15 | |
| | 5.3 | Number of Digits to Report | 16 |
| | 5.4 | Significance Level and Confidence Level | 17 |
| | 5.5 | Descriptive Statistics Values to Calculate | 17 |
| | 5.6 | Derived Variables | 17 |
| 6. | SAN | MPLE SIZE | 18 |
| 7. | STA | ATISTICAL METHODOLOGY | 19 |
| | 7.1 | Disposition of Subjects | 19 |
| | 7.2 | Demographic and Other Baseline Characteristics | 19 |
| | 7.3 | Medical History and Allergic History | 19 |
| | 71 | Prior and Concomitant Medications | 19 |

| 7.5 | Study | Drug Exposure and Treatment Compliance | 20 |
|-----|---------|-----------------------------------------------------|----|
| 7.6 | Statist | ical/Analytical issues | 20 |
| - | 7.6.1 | Adjustments of Covariates | 20 |
| | 7.6.2 | Handling of Dropouts or Missing Data | 20 |
| | 7.6.3 | Interim Analyses and Data Monitoring | 20 |
| | 7.6.4 | Multicentre Studies | 20 |
| | 7.6.5 | Multiple Comparison/Multiplicity | 20 |
| | 7.6.6 | Use of an "Efficacy Subset" of Patients | 20 |
| | 7.6.7 | Active-Control Studies Intended to Show Equivalence | 21 |
| | 7.6.8 | Examination of Subgroups | 21 |
| | 7.6.9 | Handling of Laboratory Test Values | 21 |
| 7.7 | Pharm | acokinetic Assessments | 21 |
| | 7.7.1 | Analysis of Individual Plasma Concentrations | 21 |
| | 7.7.2 | Analysis of Pharmacokinetic Parameters | 22 |
| | 7.7.3 | Analysis of Dose Proportionality | 22 |
| | 7.7.4 | Analysis of Food Effect | 23 |
| | 7.7.5 | Analysis of Racial Differences | 24 |
| | 7.7.6 | Analysis of Difference by Adding Thickener | 24 |
| | 7.7.7 | Analysis of Steady State | 25 |
| | 7.7.8 | Analysis of Linearity | 25 |
| | 7.7.9 | Analysis of Accumulation | 26 |
| 7.8 | Safety | Assessments | 27 |
| | 7.8.1 | Adverse Events | 27 |
| | 7.8.2 | Laboratory Tests | 27 |
| | 7.8.3 | Vital Signs | 28 |
| | 7.8.4 | 12-lead ECG | 28 |
| | 7.8.5 | Physical Examinations | 29 |

#### Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation.

| | 7.8.6 | Withdrawals | 29 |
|----|-------|------------------------------------------|----|
| | 7.8.7 | Sensory Tests | 29 |
| | 7.8.8 | Other Safety Assessments | 29 |
| 8. | | FROM THE PROTOCOL | |
| | | T SUMMARISED OR PRESENTED | |
| | | CES | |
| | | IONS | |
| | | , TABLES AND FIGURES | |
| | | gs | |
| | | S | |
| | | es | |
| 13 | | HISTORY FOR SAP AMENDMENTS | |
| | | – PHARMACOKINETIC PARAMETER CALCULATIONS | |

#### Abbreviations

AE : adverse event

ANOVA: analysis of variance

 $\alpha$ : intercept of regression line

β : slope of regression line

BLQ : below limit of quantification

BMI : body mass index

CI : confidence interval

CV : coefficient of variation

DBL: database lock

DP : decimal places

ECG: electrocardiogram

IAO : International Agreed Order

IMP : investigational medicinal product

LLOO: lower limit of quantification

LF : linearity factor

LOQ: limit of quantification

LSmeans: least squares means

MedDRA: Medical Dictionary for Regulatory Activities

NC: not calculated

PK: pharmacokinetics

PP : per protocol

PT : preferred term

QC : quality control

r : Pearson's correlation coefficient

RA: ratio of accumulation

SAP : statistical analysis plan

SAE : serious adverse event

SD : standard deviation

SOC : system organ class

TEAE : treatment emergent adverse event

WHO-DD: World Health Organization Drug Dictionary

| Parameters | Unit | Definitions |
|---|---|---|
| AUC <sub>0-8h</sub><br>AUC <sub>0-12h</sub><br>AUC <sub>0-24h</sub> | h•ng/mL | Area under the plasma concentration-time curve from 0 to 8, 12 or 24 h |
| AUC <sub>0-last</sub> | h•ng/mL | Area under the plasma concentration-time curve from zero up to the last quantifiable concentration time point |
| AUC₀-∞ | h•ng/mL | Area under the plasma concentration-time curve from zero up to infinity with extrapolation of the terminal phase |
| AUC <sub>0-τ</sub> | h•ng/mL | Area under the plasma concentration-time curve over a dosing interval |
| AUC% <sub>ex</sub> | % | Area under the plasma concentration-time curve extrapolated from the last quantifiable concentration time point to infinity in % of the total $AUC_{0-\infty}$ |
| C <sub>max</sub> | ng/mL | Maximum plasma concentration |
| Clast | ng/mL | Last quantifiable concentration |
| CL/F | L/h | Apparent total clearance |
| C <sub>trough</sub> | ng/mL | Minimum plasma concentration |
| $\lambda_{z}$ | /h | Terminal elimination rate constant |
| Lower limited of $\lambda_z$ | h | Lower data point used for the estimation of $\lambda_z$ |
| MRT <sub>0-∞</sub> | h | Mean residence time from zero up to infinity with extrapolation of the terminal phase |
| MRT <sub>ss</sub> | h | Mean residence time at steady state |
| Number of $\lambda_z$ points | | Number of data point used for the estimation of $\lambda_z$ |
| t <sub>1/2</sub> | h | Terminal elimination half-life |
| t <sub>max</sub> | h | Time to reach the maximum plasma concentration |
| Upper limited of $\lambda_z$ | h | Upper data point used for the estimation of $\lambda_z$ |
| V <sub>ss</sub> /F | L | Apparent distribution volume at steady state |
| V <sub>z</sub> /F | L | Apparent distribution volume at the elimination phase |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) is based on the final protocol dated 2 July 2018. The plan covers statistical analysis plan, tabulations and listings of pharmacokinetic (PK) and safety data to assess the pharmacokinetics, safety, and tolerability of single and multiple doses of edaravone solution and suspension in healthy adult males. Holter ECG analysis with the related section of 2.1.2 and 2.2.3 will be performed in a separate ECG SAP.

The SAP is prepared by The statistical analyses and production of the outputs described in the SAP will be conducted and QC checked by Data Science Department, using SAS® 9.3 or a later version. The final analyses and outputs will be approved by Mitsubishi Tanabe Pharma Corporation.

#### 1.1 Study Design

Phase of the study: I

Type of study: Clinical pharmacology study

This study will be performed using a placebo-controlled, randomized, single-blind design, and consists of Part 1 (single-dose study) and Part 2 (multiple-dose study).

The flow of cohort transition in this study is shown in Figure 1. Except in Cohorts S3-1 and S3-2, no subjects will be administered the study drug in multiple cohorts.



Cohort No., Dose /day, (fasting /after meal), race, randomization rate (E:edaravone, P:Placebo)
\* Temporary dose, Dose will be decided based on PK and safety data in the previous cohort.

Figure 1 Cohort Transition Flow

#### 1.2 Schedule of Study Procedures

Study assessments are summarized in the Test/Observation Schedule.

> Mitsubishi Tanabe Pharma Corporation. Statistical Analysis Plan

(1) Part 1: Single-dose study

At least a 4-day (≥96 hours) washout period will be required between doses of S3-1 and S3-2. The end-of-study assessment in S3-1 can be replaced by the hospitalization assessment in S3-2.

| Study period | Screening | | | | | | | Hospitalization | ization | | | | | | | | End-of-study<br>assessment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Ned | -30 to -2 | a) | | | | | | 1 | Section 1985. | | | | | | 2 | 8 | 8 (±2) |
| Time point | | 5 | Pre-dose | 0 | 0.25 | 0.5 | | 1.5 | 2 | 3 | 4 6 | 8 | 12 | 24 | 36 | 48 | |
| Hospitalization | Visiting | | | | | H | | 1 | + | + | $\frac{1}{1}$ | $\prod$ | $\parallel$ | | | | Visiting |
| Meals (B, breakfast;<br>L, lunch; S, supper) | В <sup>2)</sup> х | B <sup>-t,</sup> ×<br>L, S O<br>Fasting from<br>11:00 p.m. | B <sup>3)</sup><br>×/O | | | | | | L, S O | | | | | | 0 | B only | B <sup>2)</sup> × |
| Informed consent | × | | | | | | | | | - | 1 | | | _ | | | |
| Medical history,<br>complications,<br>demographic<br>characteristics | × | | | | | . : | | | | | | | | _ | | | |
| Inclusion/exclusion criteria | × | × | × | | | | | | | - | | | _ | | | | |
| Study drug<br>administration | | | | X <sub>3</sub> | | | | | · | | | | | | | | |
| Serological test | × | | | | | | | | - 1 | | | 4 | _ | | | | |
| Drug and alcohol abuse screening | × | × | | | | | | | | | | | | | | | |
| Height, body weight, BMI | × | × | | | | | | | | | | | | | | | × |
| Physical<br>examination <sup>5)</sup> | × | × | × | | | | × | | | × | <u>×</u> | | <u>×</u> | × | | × | × |
| Vital signs | × | × | × | | | | × | | | × | × | | × | × | | × | × |
| 12-lead ECG" | × | × | X | | | | × | | | 4 | | - | × <br>- | × | - | × | × |
| Holter ECG" | | | × | | × | × | $\prec$ | $\stackrel{ }{\times}$ | × | | ^<br> <br> | <u> </u> | <u> </u> | <b>*</b> } | $\stackrel{A}{+}$ | × | > |
| Laboratory tests" | × | × | | | | | 1 | 1 | | + | 1 | | - | <u>{</u> | | | <b>\</b> |
| AEs | | | | $\bigvee$ | | | | $\parallel$ | | $\ $ | $\ $ | $\prod$ | $\parallel$ | $\prod$ | | | N |
| Concomitant medications | From Day<br>-7 | | | | | | | | | | H | | | | | | |
| Blood sampling for plasma drug concentration | | | × | - | × | × | × | × | × | | × × | <u>×</u> | <u>×</u> | × | × | × | |
| incasulation 10.00 | 0.0 | | | | | | 1 | l | | 1 | ł | | | | | | |

Hospitalization at around 9:00 a m. Subjects will skip breakfast after the completion of tests. 7

## Mitsubishi Tanabe Pharma Corporation. Statistical Analysis Plan

Protocol No. MT-1186-J01 Date: 9 October, 2018

- Subjects in Cohorts S1, S2, S3-1, S4, S5, S6, and S7 will skip breakfast (administration under fasting conditions). Subjects in Cohort S3-2 will have tests first. After having breakfast, they will be given the study drug (administration 30 minutes after a meal). 3
  - Height will be measured at screening only. Body weight will be measured at screening, hospitalization, and end-of-study assessments. BMI will be calculated at screening and hospitalization assessment. 4
- A physical examination, vital signs (systolic and diastolic blood pressure, pulse rate, and body temperature), and a 12-lead ECG will be assessed at the following time points: screening, at hospitalization, pre-dose, 1, 3, 6, and 12 hours post-dose, before breakfast on Days 2 and 3, and end-of-study assessment.

  Holter ECG data will be recorded in Cohorts S4, S5, and S6 at the following time points: 45, 30, and 15 minutes pre-dose, 15 and 30 minutes post-dose and 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 3
- 6
  - Laboratory tests (hematology, biochemistry, coagulation test, and urinalysis): The hospitalization assessment will be performed based on results that can be confirmed within the same and 48 hours post-dose. 6
    - day. The laboratory tests will be performed at screening, hospitalization assessment, before breakfast on Day 2, and end-of-study assessment.
      - Blood will be drawn at pre-dose, 15 and 30 minutes post-dose and 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose for drug concentration measurement.

Mitsubishi Tanabe Pharma Corporation. Statistical Analysis Plan

[For 5-day administration] (2) Part 2: Multiple-dose study

| Study period | Screening | | | | | Hospitalization | | | | | End-of-study<br>assessment |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | -30 to -2 | F | | | 7 | e | 7 | 2 | 9 | 1 | 12 (±2) |
| | | At<br>hospitaliza<br>fion | Pre-dose | Post-dose | | | | Day of last<br>dose | | | |
| Hospitalization | Visiting | | | | | | | | | 1 | Visiting |
| Meals (B, breakfast, L, lunch, S, supper) | В <sup>2)</sup> х | B <sup>21</sup> ×<br>L, S O<br>Fasting<br>from 11:00<br>p.m. | | B, L, S <sup>10)</sup> | O <sup>10)</sup> | O <sup>10)</sup> | O 10) | O <sup>10)</sup> | 0 | B only | В <sup>2)</sup> х |
| Informed consent | × | | | | | | | | | | |
| Medical history, complications, demographic characteristics | × | | | | | | | | | | |
| Inclusion/exclusion criteria | × | × | × | | | Ş | Į. | 7 | | | |
| Study drug administration | | | | ,<br>X | £ | ķ | ķ | × | | | |
| Serological test | × | | | | | | | | | | |
| Drug and alcohol abuse screening | × | × | | | | | · | | | | |
| Height, body weight, BMI <sup>5)</sup> | × | × | | | | | | | | | × |
| Physical examination <sup>6)</sup> | × | × | × | × | × | × | × | × | × | × | × |
| Vital signs <sup>8)</sup> | × | × | × | × | × | × | × | × | × | × | × |
| 124ead ECG <sup>6)</sup> | × | × | × | × | × | × | × | × | × | × | × |
| Sensory tests <sup>()</sup> | | × | | | | | | | × | | |
| Laboratory tests <sup>8)</sup> | × | × | | | | × | | | × | | × |
| AEs | | | | V | | | | | | | |
| Concomitant medications | From Day – | | | | | | | | | | $\uparrow$ |
| Blood sampling for plasma drug | | | | | | | | | | ^ | |
| concentration measurement <sup>a)</sup> | | | , | | ŀ | | | | | | |
| m > OOO parton of confirmation of one | 200 | | | | | | | | | | |

Hospitalization at around 9:00 a.m. Subjects will skip be study site. They can have breakfast after the completion of tests. Subjects will skip breakfast and visit the study site. They can have breakfast after the study drug will be administered in the morning only.) Administration in the morning only (Even in the twice-daily administration regimen, the study drug will be administered in the morning only.) 963

# Protocol No. MT-1186-J01

Date: 9 October, 2018

Mitsubishi Tanabe Pharma Corporation. Statistical Analysis Plan

- in the morning and before bedtime (12 hours after the morning dose). For morning administration under fasting conditions, breakfast will be 30 minutes, 1 hour or 90 Once- or twice-daily administration. For once-daily administration, the study drug will be given in the morning. For twice-daily administration, the study drug will be given minutes after administration, or not eaten. 4
  - Height will be measured at screening only. Body weight will be measured at screening, hospitalization, and end-of-study assessments. BMI will be calculated at screening and the hospitalization assessment. 2
- A physical examination, vital signs (systolic and diastolic blood pressure, pulse rate, and body temperature), and a 12-lead ECG will be assessed at the following time points: screening, at hospitalization, pre-morning dose, 1, 3, 6, and 12 hours post-dose on Days 1 to 5, before breakfast on Days 6 and 7, and end-of-study assessment. 6
  - Sensory tests will be performed at hospitalization assessment and before breakfast on Day 6.
  - Laboratory tests (hematology, biochemistry, coagulation test, and urinalysis): The hospitalization assessment will be performed based on results that can be confirmed within the same day. Laboratory tests will be performed at screening, hospitalization assessment, on Days 3 and 6, and end-of-study assessment. 68
    - Day 1: Prior to administration in the morning (first dose), 15 and 30 minutes post-dose, and 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose 3lood sampling for drug concentration measurement: 6
- Day 5: Prior to the last dose (administration in the morning), 15 and 30 minutes post-dose, and 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose Day 2: Prior to administration in the morning (about 24 hours after the first dose) Days 3 and 4: Prior to administration in the morning
  - Day 6: 24 hours after the last dose Day 7: 48 hours after the last dose
- Breakfast will be 30 minutes, 1 hour or 90 minutes after administration, or not eaten. 10

#### 2. STUDY OBJECTIVE(S) AND ENDPOINTS

#### 2.1 Study Objective(s)

#### 2.1.1 Primary Objective(s)

The primary objective of this study is to evaluate the PK, safety, and tolerability of single and multiple doses of edaravone solution and suspension in healthy adult males.

#### 2.1.2 Secondary Objectives

The secondary objectives of this study is to confirm the PK profiles of a single dose of edaravone suspension in different races, fed/fasted conditions, and different drug dissolution profiles and to collect ECG data to evaluate QTcF prolongation and proarrhythmic potential for edaravone.

#### 2.2 Endpoints

#### 2.2.1 Safety Endpoints

- (1) AEs and ADRs
- (2) 12-lead ECG
- (3) Vital signs
- (4) Laboratory tests
- (5) Sensory tests

#### 2.2.2 Pharmacokinetic Endpoints

(1) Plasma drug concentrations
Unchanged edaravone, sulfate conjugate, and glucuronide conjugate

(2) PK parameters

AUC<sub>0-last</sub>, AUC<sub>0-8h</sub>, AUC<sub>0-12h</sub>, AUC<sub>0-24h</sub>, AUC<sub>0- $\infty$ </sub>, C<sub>max</sub>, C<sub>trough</sub>, t<sub>max</sub>, t<sub>1/2</sub>,  $\lambda_z$ , MRT\*, CL/F\*, V<sub>z</sub>/F\*, and V<sub>ss</sub>/F\* (\*: calculated for unchanged edaravone only)

#### 2.2.3 Pharmacodynamic Endpoints

Heart rate, QTcF, PR interval, QT interval, RR interval, and QRS interval from Holter ECG

#### 3. PLANNED ANALYSES

This study was planned to examine the pharmacokinetics (PK), safety, and tolerability of oral administration of edaravone.

The statistical analyses will be performed after database lock(DBL). Interim analysis will not be carried out.

#### 4. ANALYSIS POPULATION(S)

The definitions of the analysis sets are provided below. The detailed handling of subjects will be determined by the sponsor, by the time of the data lock.

- (1) Safety analysis set

  The safety analysis set will consist of all subjects who received at least 1 dose of the study drug.
- (2) PK analysis set

  The PK analysis set will consist of all subjects who received at least 1 dose of the study drug and had evaluable PK data.

For cases that subjects were not adopted in the PK analysis set, all PK data will be rejected and no parameters will be calculated. Furthermore, for cases that subjects adopted in the PK analysis set and partial data not being adopted, PK parameters will be calculated from only the adopted data.

The acceptance or rejection of each analysis population will be treated based on the results of the data review meeting on as follows.

Safety analysis set: No subject is excluded from analysis.

PK analysis set: No subject is excluded from analysis.

#### 5. GENERAL CONSIDERATIONS

In the single-dose and multiple-dose studies, data collected at each dose of each cohort, and the corresponding pooled data of the placebo group will be summarized.

#### 5.1 Subjects Composition

The dose, dosing regimen, and duration of administration for each cohort of Part 1 and 2 are shown in the tables below.

Except in Cohorts S3-1 and S3-2, no subjects will be administered the study drug in multiple cohorts.

#### (1) Part 1 (single-dose study)

A single oral dose of the study drug will be given to subjects under fasting conditions in the morning or 30 minutes after breakfast. In Cohort S3-2, subjects in Cohort S3-1 will be given the same study drug that is allocated in Cohort S3-1 in a single oral dose after at least a 4-day washout period.

Table. Dose, Dosing Regimen, and Duration (Single-dose study [Part 1])

| Cohort | Dose | Condition of | Race | Duration | No. of s | ubjects |
|---|---|---|---|---|---|---|
| | | administration | | | Edaravone | Placebo |
| S1 | 60 mg | | | 1 day | 6 | 2 |
| S2 | 120 mg <sup>1)</sup> | Fasting | | 1 day | 6 | 2 |
| S3-1 | 200 mg <sup>1)</sup> | | Tomonogo | 1 day | 6 | 2 |
| S3-2 | ]200 mg | After a meal | Japanese | 1 day | | |
| S4 <sup>1)</sup> | 300 mg <sup>1)</sup> | | } | 1 day | 6 | 2 |
| S5 | 300 mg <sup>1)</sup> | Fasting | | 1 day | 6 | 2 |
| S6 | 30 mg | | | 1 day | 6 | 2 |
| S7 <sup>2)</sup> | 200 mg <sup>1)</sup> | ] | Caucasian | 1 day | 6 | 2 |

<sup>1)</sup> For Cohort S4, polyvinyl alcohol and xanthan gum will be used as vehicles. Cohort S4 can be started using same timing as Cohort S3-2.

#### (2) Part 2 (multiple-dose study)

A once-daily oral dose of the study drug will be given to subjects 30 minutes before breakfast. (For Day 1 and Day 5 [day of the last dose], an oral dose of the study drug will be administered 30 minutes before breakfast only.)

Table. Dose, Dosing Regimen, and Duration (Multiple-dose study [Part 2])

| Cohort | Dose | Frequency of | Duration | No. of s | ubjects |
|--------|--------|----------------|----------|-----------|---------|
| | | administration | | Edaravone | Placebo |
| M1 | 120 mg | Once daily | 5 days | 6 | 3 |
| M2 | 200 mg | Once daily | 5 days | 6 | 3 |

#### 5.2 Analysis Time Window for Visits

In Part 1 (single-dose study), analysis time windows for blood sampling for PK measurements are as follows.

| Pre-dose | before dosing |
|---|---|
| 0.25 h, 0.5 h, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h and 12 h after | Scheduled time ± 5 minutes |
| dosing | |

<sup>2)</sup> The dose in Cohort S7 will be the same as that in Cohorts S3-1 and S3-2. Cohort S7 can be started using the same timing as Cohort S3-1.

| 24 h, 36 h and 48 h after dosing | Scheduled time ± 15 minutes |
|----------------------------------|-----------------------------|

In Part 2 (multiple-dose study), analysis time windows for blood sampling for PK measurements are as follows.

| Pre-dose (Day 1 to Day 5) | before first dosing |
|---|---|
| 0.25 h, 0.5 h, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h and 12 h after first dosing | Scheduled time ± 5 minutes |
| Pre-dose (Day 2: Day 1 24 h after first dosing) | Scheduled time - 15 minutes |
| Pre-dose (Day 3 to Day 4) | Scheduled time - 15 minutes |
| Pre-dose (Day 5: before last dosing) | Scheduled time - 15 minutes |
| 0.25 h, 0.5 h, 1 h, 1.5 h, 2 h, 4 h, 6 h, 8 h and 12 h after last dosing (Day 5) | Scheduled time ± 5 minutes |
| 24 h (Day 6) after last dosing | Scheduled time ± 15 minutes |
| 48 h (Day 7) after last dosing | Scheduled time ± 15 minutes |

Analysis time windows for safety evaluation are as follows.

| Screening (Day -30 to Day -2) | Not specified* |
|---|---|
| Hospitalization (Day -1) | Not specified* |
| Before dosing (Day 1 to Day 5) | Before dosing time |
| 1 h, 3 h, 6 h, and 12 h after dosing (Day 2 to Day 4) 1 h, 3 h, 6 h, 12 h, 24 h, and 48 h after dosing (Day 1, Day 5) | Not specified* |
| Follow-up (Day 8 ± 2days, Day 12 ± 2days) | Not specified* |

<sup>\*</sup> By-visit safety analysis will be summarized by the nominal visit number. Assessment taken outside of protocol allowable windows such as end of study assessment (+2) will be displayed according to the case report form assessment recorded by the investigator.

If a re-examination was performed except Follow-up or later, it will be evaluated at the applicable visit.

#### 5.3 Number of Digits to Report

Statistical analysis variables, statistics to be calculated and number of digits to report are as follows.

| Laboratory tests Physical examinations Standard 12-Lead ECG | Mean, SD, median | Report to one extra digit plus the determined/specified digits |
|---|---|---|
| | Minimum, maximum | Report to the determined/specified digits |
| Pharmacokinetics | Mean, SD, minimum, median,<br>maximum, SE, geometric mean,<br>LSmeans, geometric LSmeans, CI | Report to the determined/specified digits |

| | Degree of freedom | Integer If degree of freedom is adjusted by Kenward-Roger approximation, rounded |
|---|---|---|
| | Sum of squares, Mean square | off to one decimal place. To the 4 decimal places |
| | α, β, r | 4 significant digits |
| | F-value | To the 2 decimal places the following also applies: if F-value<0.01, displayed "F<0.01". |
| | p-value | To the 4 decimal places the following also applies: if p-value<0.0001, displayed "p<0.0001". |
| General information | Number of subjects, number of valid observations, number of events, number of cases | Integer |
| | CV%, geometric CV%,<br>Percentages (%) | To the first decimal place |
| | Ratio | To the 3 decimal places |

#### 5.4 Significance Level and Confidence Level

The significance level of the statistical test will be 5% (two-sides). The two-sided confidence level of the confidence interval will be 95%. The two-sided confidence level for comparison between groups will be 90%.

#### 5.5 Descriptive Statistics Values to Calculate

Where appropriate, continuous variables will be summarized descriptively, using the number of observations, mean, SD, median, minimum, and maximum. Categorical variables will be summarized using frequency counts and percentages. In the single-dose and multiple-dose studies, data pooled of placebo groups in the data collected at each dose of each cohort will be summarized.

#### 5.6 Derived Variables

#### (1) Definition(s) of baseline(s)

The baseline of vital signs and 12-lead ECG is the final evaluable value obtained before IMP administration on Day 1.

The baseline of clinical laboratory values will be the value obtained on Day -1.

Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation.

#### (2) Age at informed consent

Age (years) = Year of informed consent - Year of birth

Subtract 1 from the age (years) calculated above, if [Month of informed consent < Month of birth] or [Month of informed consent = Month of birth AND Day of informed consent < Day of birth].

#### (3) BMI

BMI = Body weight (kg) / height (m) $^2$  (rounded to one decimal place)

Height will be the value obtained at screening.

Body weight will be the value obtained at Day -1.

#### (4) eGFR

eGFR (mL/min/1.73m<sup>2</sup>) = 194 × creatinine (mg/dL)<sup>-1 094</sup> × Age (years)<sup>-0 287</sup>

Age will be the value obtained at informed consent.

However, in cohort S7, GFR will be calculated by MDRD equation.

eGFR (mL/min/1.73m<sup>2</sup>) = 175 × creatinine (mg/dL)<sup>-1</sup> 154 × Age (years)<sup>-0</sup> 203

#### (5) Adverse events

The MedDRA/J (version 20.0 or a later version) will be used as a unified dictionary in the assessment of AEs.

#### (6) Adverse reactions

Adverse reactions are defined as AEs that are determined to have a "Reasonable Possibility" of causal relationship to the IMP.

#### 6. SAMPLE SIZE

A total of 74 subjects

Part 1 (single-dose study): 56 subjects

(8 subjects per cohort: 6 subjects in the edaravone group and 2

subjects in the placebo group)

Part 2 (multiple-dose study): 18 subjects

(9 subjects per cohort: 6 subjects in the edaravone group and 3

subjects in the placebo group)

#### 7. STATISTICAL METHODOLOGY

#### 7.1 Disposition of Subjects

Disposition of subjects will be listed.

- Number and percent of subjects completed protocol scheduled visits will be presented.
- > Subjects' status for each cohort will be summarized wherever applicable. Subjects who discontinued in each cohort will be summarized by reasons for discontinuation.

#### 7.2 Demographic and Other Baseline Characteristics

All demographic and other baseline characteristics will be listed.

For safety analysis set, all demographic and other baseline characteristics will be summarized. For countable values, frequency and percentage will be reported. For metric values, descriptive statistics values (number of subjects, mean, SD, minimum, median, and maximum) will be calculated.

Table. Variables related to demographic and other baseline characteristics

| Category | Variable | Data format |
|------------|---------------------------------------------|-------------|
| Subject | Sex (male, female): display without female | Binary |
| background | Age at consent acquisition (years) | Metric |
| | Height (cm) | Metric |
| | Body weight (kg) on Day -1 | Metric |
| | BMI on Day -1 | Metric |
| | Race | Binary |
| | Medical history | Binary |
| | Complications | Binary |
| | Allergic History (including drug allergies) | Binary |
| | Drinking status, Stratified into 2: | Dinama |
| | 'NEVER' (No) vs. otherwise (Yes). | Binary |
| | Smoking status, Stratified into 2: | Dinami |
| | 'NEVER' (No) vs. otherwise (Yes). | Binary |

#### 7.3 Medical History and Allergic History

All medical history and allergic history data will be listed.

#### 7.4 Prior and Concomitant Medications

All medications data will be listed.

All medications data will be coded according to the latest version of WHO-DD and Anatomical Therapeutic Chemistry (ATC) classification, and will be summarized by each cohort. Prior and

Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation.

concomitant medications will be summarized separately. Incidence tables will be summarized with ATC Level 2 code, text and Drug Code, Drug Name.

Prior medication is any medication that was stopped prior to the first intake of IMP. Concomitant medication is any medication that is on-going at the time of the first dose or started after the first intake of IMP. Concomitant medications with an incomplete start date but that are still ongoing at the end of the study will be considered as concomitant medications.

Regarding timing of concomitant medications used in cohorts S3-1 and S3-2, concomitant medications used before dose of S3-2 is taken as S3-1, and concomitant medications used after dose of S3-2 is taken as S3-2. If there is no record of the used time of the concomitant medications used on the same day as the dosing day of S3-2 is taken as S3-2.

#### 7.5 Study Drug Exposure and Treatment Compliance

All exposure and compliance data will be listed.

#### 7.6 Statistical/Analytical issues

#### 7.6.1 Adjustments of Covariates

Adjustments of covariates will not be performed.

#### 7.6.2 Handling of Dropouts or Missing Data

Missing data, such as rejected values, will not be imputed.

#### 7.6.3 Interim Analyses and Data Monitoring

Not applicable in the study.

#### 7.6.4 Multicentre Studies

Not applicable in the study.

#### 7.6.5 Multiple Comparison/Multiplicity

Adjustments of multiplicity will not be performed.

#### 7.6.6 Use of an "Efficacy Subset" of Patients

Not applicable in the study.

#### 7.6.7 Active-Control Studies Intended to Show Equivalence

Not applicable in the study.

#### 7.6.8 Examination of Subgroups

Not applicable in the study.

#### 7.6.9 Handling of Laboratory Test Values

In the case of clinical laboratory test values including equality and inequality sign, exclude equality and inequality sign and use for summarized.

#### 7.7 Pharmacokinetic Assessments

The Pharmacokinetics parameters of unchanged edaravone, sulfate conjugate, and glucuronide conjugate will be calculated by Non-compartmental analysis using Phoenix® WinNonlin® 6.3 or a later version Software. The time used to calculate the pharmacokinetic parameters will be the actual time (rounded to two decimal places) with the time of the IMP administration taken as 0.00 hours. When the same parameter has Observed and Predicted values, Observed value will be adopted. In addition, the concentration below the quantitation limit (BLQ) will be considered as a numerical value of 0 and calculation will be performed.

#### 7.7.1 Analysis of Individual Plasma Concentrations

All measured plasma concentrations will be listed.

Plasma concentrations will be summarized at each scheduled sampling time point by each cohort. The following descriptive statistics will be calculated: N (number of subjects), n (number of valid observations), arithmetic mean, SD, CV%, minimum, median, maximum, geometric mean and geometric CV%. Nominal sampling times will be displayed in the summary. For the calculation of the descriptive statistics other than geometric mean and geometric CV%, concentration values reported as BLQ will be set to 0. For the calculation of the geometric mean and geometric CV%, concentration values reported as BLQ will be set to ½ of LLOQ.

CV% and Geometric CV% will be calculated as follows:

$$CV\% = \frac{SD}{arithmetic\ mean} \times 100$$

Geometric CV% = 
$$\left[\exp(\sigma^2) - 1\right]^{1/2} \times 100$$

where  $\sigma$  represents the SD computed on the natural logarithmic transformed concentrations.

To visualize the concentration-time profiles of each cohort, the following plots will be produced in linear and semi-logarithmic scales:

- 1. Individual subject concentration-time plot overlaid in one graph by cohort.
- 2. Mean concentration-time plot for each cohort overlaid in one graph.

In the summary tables, arithmetic mean, SD, minimum, median, maximum and geometric mean will be presented with the number of significant digits which individual concentrations are reported. In addition, CV%, and geometric CV% will be presented with 1 decimal place.

#### 7.7.2 Analysis of Pharmacokinetic Parameters

All PK parameters will be listed.

The PK parameters will be summarized by each cohort. The following descriptive statistics will be calculated: N (number of subjects), n (number of valid observations), arithmetic mean, SD, CV%, minimum, median, maximum, geometric mean and geometric CV%.

For the descriptive statistics, the minimum and maximum will be presented according to following requirement:

- t<sub>max</sub>: will be presented with 2 decimal places.
- $C_{max}$ ,  $C_{max}/D$ ,  $C_{max}$ \*kg: will be presented with the number of significant digits they are reported with.
- Number of  $\lambda_z$  points: will be presented with integer.
- Other PK parameters: will be presented with a fixed number of decimal places for each parameter. The number of decimal places is 2 decimal places corresponding to having 3 significant digits at the minimum by analyte.

Mean, SD, median and geometric mean will be presented with the number of decimals as follows.

- $C_{max}$ ,  $C_{max}$ /D,  $C_{max}$ \*kg: will be presented with the number of significant digits they are reported with.
- Other PK parameters: will be presented with 2 decimal places.

CV% and geometric CV% will be presented with 1 decimal place.

#### 7.7.3 Analysis of Dose Proportionality

In Part 1 (single-dose study), dose proportionality test on  $C_{max}$ ,  $AUC_{0-8h}$ ,  $AUC_{0-last}$  and  $AUC_{0-\infty}$  (except for Cohort S3-2 and S7) of unchanged edaravone, sulfate conjugate, and glucuronide conjugate will be performed with log-transformed doses by power model analysis. In this model,  $Y=aX^{\beta}$  (Y:plasma pharmacokinetic parameter,X:dose) is also described as a simple regression model,  $ln(Y)=\alpha+\beta\times ln(X)$  [ $\alpha=ln(a)$ ] when both sides of the formula are log-transformed. If confirm the suitability by Lack-of-Fit test, and the two-sided 95% confidence interval of the slope ( $\beta$ ) includes "1", the parameter will be considered dose-proportional.

Adequacy of the power model will be measured by Lack-of-Fit test. Insignificant Lack-of-Fit test indicates that the model is adequate to confirm linearity.

If dose-proportionality or linear regression fit is not demonstrated for any of the pharmacokinetic parameters in the range of 5 dose groups (30, 60, 120, 200, and 300 mg), dose-proportionality will be examined with smaller dose ranges by reducing one dose each from the highest (300 mg) up to the smallest range with 3 lowest doses (30, 60, and 120 mg) to make an exploratory investigation of the proportional dose range. Furthermore, in addition to the range of the above dose group, the dose groups (120, 200, and 300 mg) of only administration of suspension, and the dose groups (120, 200, and 300 mg, except for Cohort S4), and (30, and 60 mg) of 2 different formulation of the same viscosity will be also performed. Incidentally, in the 2 dose group will not be performed the Lack-of-Fit test.

#### SAS Code



Log-log scatter plot of regression lines and their two-sided 95% confidence intervals will be created for all cohorts (except for Cohort S3-2 and S7) to investigate the correlation between the pharmacokinetic parameters and dose, with dose on the horizontal axis and parameters on the vertical axis on Log-log plots, whether or not the adequacy of the power model is demonstrated.

Schematic Box-and-Whisker plots at  $C_{max}/D$ ,  $AUC_{0-8h}/D$ ,  $AUC_{0-last}/D$  and  $AUC_{0-\infty}/D$  will be created, juxtaposing on the same graph by each cohort.

#### 7.7.4 Analysis of Food Effect

In Cohorts S3-1 and S3-2, mixed effect model of repeated measurements for log-transformed  $C_{max}$ ,  $AUC_{0-last}$  and  $AUC_{0-\infty}$  of unchanged edaravone, sulfate conjugate, and glucuronide conjugate will be performed with cohorts, and subjects as a factor. The differences in LSmeans and their two-sided 90% confidence intervals will be calculated.

LSmeans and their two-sided 90% confidence intervals for differences between fasted and fed treatments will be calculated by each cohort. Exponentially transformed values as ratio of geometric LSmeans will be presented for these analyses.

CS (Compound Symmetry) will be presupposed for structure of variance-covariance considering correlation among cohorts. Kenward-Roger approximation will be used for adjustment of degree of freedom.

#### SAS Code



Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation.



Schematic Box-and-Whisker plots juxtaposing the above pharmacokinetic parameters at fasted and fed administration will be created on the same graph.

Ratio of geometric LSmeans of  $C_{max}$ ,  $AUC_{0-last}$  and  $AUC_{0-\infty}$  between dosing conditions (fed/fasted) and its two-sided 90% confidence interval will be presented with forest plots on the same graph.

#### 7.7.5 Analysis of Racial Differences

In Cohorts S3-1 and S7, mixed effect model for log-transformed  $C_{max}*kg$ ,  $AUC_{0-last}*kg$ ,  $AUC_{0-last}$  and  $AUC_{0-\infty}$  of unchanged edaravone, sulfate conjugate, and glucuronide conjugate will be performed with cohorts, and subjects as a factor. The differences in LSmeans and their two-sided 90% confidence intervals will be calculated.

LSmeans and their two-sided 90% confidence intervals for racial differences will be calculated by each cohort. Exponentially transformed values as ratio of geometric LSmeans will be presented for these analyses.

Kenward-Roger approximation will be used for adjustment of degree of freedom.

SAS Code



Schematic Box-and-Whisker plots at  $C_{max}$ \*kg,  $AUC_{0-last}$ \*kg,  $AUC_{0-\omega}$ \*kg,  $C_{max}$ ,  $AUC_{0-last}$  and  $AUC_{0-\omega}$  will be created, juxtaposing on the same graph by each cohort.

#### 7.7.6 Analysis of Difference by Adding Thickener

In Cohorts S4 and S5, mixed effect model for log-transformed  $C_{max}$ ,  $AUC_{0-last}$  and  $AUC_{0-\infty}$  of unchanged edaravone, sulfate conjugate, and glucuronide conjugate will be performed with cohorts, and subjects as a factor. The differences in LSmeans and their two-sided 90% confidence intervals will be calculated.

LSmeans and their two-sided 90% confidence intervals for difference between presence or absence of thickener will be calculated by each cohort. Exponentially transformed values as ratio of geometric LSmeans will be presented for these analyses.

Kenward-Roger approximation will be used for adjustment of degree of freedom.

#### SAS Code



Schematic Box-and-Whisker plots at  $C_{max}$ ,  $AUC_{0-last}$  and  $AUC_{0-\infty}$  will be created, juxtaposing on the same graph by each cohort.

#### 7.7.7 Analysis of Steady State

In Part 2 (multiple-dose study), the ratio of the C<sub>trough</sub> (plasma concentration at the end of the dosing interval) of unchanged edaravone, sulfate conjugate, and glucuronide conjugate for each day of dosing to those after the last dose (C<sub>trough,DayX</sub> / C<sub>trough,ss</sub>) will be calculated for each subject, and descriptive statistics, in addition to it, geometric mean and their two-sided 95% confidence intervals will be calculated by each cohort.

Profiles of means of C<sub>trough</sub> from Days 2 to 5 at Part 2 (multiple-dose study) will be created with both linear and semi-logarithmic plots.

#### 7.7.8 Analysis of Linearity

In Part 2 (multiple-dose study), mixed effect model of repeated measurements for log-transformed  $AUC_{0-\tau}$  (last dose) and  $AUC_{0-\infty}$  (first dose) of unchanged edaravone, sulfate conjugate, and glucuronide conjugate will be performed with treatment day, cohorts, and interaction with treatment day and cohorts as a factor. The differences in LSmeans and their two-sided 95% confidence intervals will be calculated.

Differences in LSmeans and their two-sided 95% confidence intervals will be calculated by each cohort. Exponentially transformed values as ratio of geometric LSmeans will be presented for these analyses.

CS (Compound Symmetry) will be presupposed for structure of variance-covariance considering correlation among treatment day. Kenward-Roger approximation will be used for adjustment of degree of freedom.

#### SAS Code





Ratio of geometric LSmeans of LF of each cohort and its two-sided 95% confidence interval will be presented with forest plots on the same graph.

#### 7.7.9 Analysis of Accumulation

In Part 2 (multiple-dose study), mixed effect model of repeated measurements for log-transformed  $AUC_{0-\tau}$  (last dose and first dose) of unchanged edaravone, sulfate conjugate, and glucuronide conjugate will be performed with treatment day, cohorts, and interaction with treatment day and cohorts as a factor. The differences in LSmeans and their two-sided 95% confidence intervals will be calculated.

Differences in LSmeans and their two-sided 95% confidence intervals will be calculated by each cohort. Exponentially transformed values as ratio of geometric LSmeans will be presented for these analyses.

CS (Compound Symmetry) will be presupposed for structure of variance-covariance considering correlation among treatment day. Kenward-Roger approximation will be used for adjustment of degree of freedom.

#### SAS Code



Ratio of geometric LSmeans of RA of each cohort and its two-sided 95% confidence interval will be presented with forest plots on the same graph.

#### 7.8 Safety Assessments

#### 7.8.1 Adverse Events

All AEs for each subject, including multiple occurrences of the same event, will be presented in full in a comprehensive listing including subject number, treatment, severity, seriousness, action taken, outcome, relationship to treatment, onset/stop date and duration. Deaths that occur during the study will be listed.

Duration of the AE and time to the AE occurrence from start of the IMP will be calculated and presented in days and time.

AE Occurrence from Start of IMP = Date/Time of Onset-Start Date/Time of Administration.

If Time is Missing, Date of Onset - Date of Administration +1.

Duration of AE = Date/Time of Resolution - Date/Time of Onset.

If Time is Missing, Date of Resolution - Date of Onset +1.

AEs which start on or after dosing that are expressed or exacerbated are defined as treatment emergent adverse events (TEAEs).

Regarding timing of adverse event occurrence in cohorts S3-1 and S3-2, adverse event occurrence before dose of S3-2 is taken as S3-1, and adverse event occurrence after dose of S3-2 is taken as S3-2. If there is no record of the occurrence time of an adverse event occurred on the same day as the dosing day of S3-2 is taken as S3-2.

The frequency and incidence of TEAEs will be summarized by System Organ Class (SOC) and Preferred Term (PT). The summary will be sorted by International Agreed Order (IAO) for SOC and alphabetical order for PT (or by frequency from the highest to the lowest).

Following summaries of TEAEs will be presented:

- Summary of AEs by SOC and PT
- > Summary of AEs by SOC, PT and severity of event
- Summary of AEs by SOC, PT and relationship to treatment

For summaries of AEs multiple occurrences of the same event within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the same event within a subject will be counted once in the maximum intensity category (severe > moderate > mild) and/or maximum drug relationship category (reasonable possibility>no reasonable possibility). If intensity or relationship is found to be missing the most severe occurrence will be imputed for that particular summary.

Proportion of subjects with any TEAE, subjects with any related TEAE, subjects with any treatment emergent SAE, and subjects with any TEAE leading to discontinuation of the study will be summarized.

#### 7.8.2 Laboratory Tests

All laboratory parameter will be listed.

Laboratory parameter values and changes from baseline, except for urinalysis will be summarized descriptively by analysis visit window.

Clinical significance of laboratory findings will be evaluated by the Investigator with respect to pre-defined clinically relevant ranges taking into account the Investigator site's normal ranges. The laboratory data will be listed in full with clinically relevant values flagged (L=Lower than normal range, H=Higher than normal range). A listing of laboratory values will be provided for subjects with any clinical significant findings.

Lab parameter values and changes from baseline will be summarized descriptively by each cohort and analysis visit window.

Shift tables will present the changes in clinically relevant categories from baseline to each scheduled post-baseline visit. The categories will be qualitative values for Urinalysis.

#### 7.8.3 Vital Signs

All vital sign data will be listed.

Vital signs (weight, systolic blood pressure, diastolic blood pressure, pulse rate, body temperature) values and changes from baseline will be summarized descriptively by analysis visit window.

The vital sign data will be listed in full with clinically relevant values flagged (L=Lower than normal range, H=Higher than normal range). A listing of vital signs will be provided for subjects with any clinical significant findings.

#### 7.8.4 12-lead ECG

All 12-lead ECG (heart rate, RR, PR, QRS, QT, QTcF, overall evaluation) parameters and findings will be listed.

12-lead ECG parameter values and changes from baseline will be summarized descriptively by analysis visit window. Overall evaluation will be summarized using frequency and percentage.

For ECGs, number and percentage of subjects meeting the criteria listed below will be presented:

- > OTcF > 500 msec at time point
- ightharpoonup QTcF > 480 msec at time point
- $\triangleright$  QTcF > 450 msec at time point
- ➤ Change from baseline in QTcF > 30 msec
- ➤ Change from baseline in QTcF > 60 msec

Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation.

The 12-lead ECG data will be listed in full with clinically relevant values flagged (L=Lower than normal range, H=Higher than normal range). A listing of 12-lead ECG parameter values will be provided for subjects with any clinical significant findings.

#### 7.8.5 Physical Examinations

All physical examinations data will be listed.

#### 7.8.6 Withdrawals

All subjects who are withdrawn from the study will be listed, and its discontinuation assessment will be excluded from summarized.

#### 7.8.7 Sensory Tests

Sensory tests (vibratory sensation) values and changes from baseline will be summarized descriptively by group and by analysis visit window.

With respect to sensory tests (numbness and staggering), a shift table of the changes from baseline will be shown by group and by analysis visit window.

With respect to sensory tests (numbness and staggering), incidence of abnormal values will be shown.

#### 7.8.8 Other Safety Assessments

Not applicable in the study.

#### 8. CHANGES FROM THE PROTOCOL

We will not summarize the numbers (occurrences) of TEAEs.

#### 9. DATA NOT SUMMARISED OR PRESENTED

Not applicable in the study.

#### 10. REFERENCES

Not applicable in the study.

#### 11. VALIDATIONS

SAS® for Windows (release 9.3 or a later version) will be used for statistical analyses.

Phoenix<sup>®</sup> WinNonlin<sup>®</sup> (release 6.3 or a later version) will be used to calculate Pharmacokinetics Parameters.

The quality of statistical results will be ensured by double programming a



#### 12. LISTINGS, TABLES AND FIGURES

#### 12.1 Listings

| No. | Title of listing | Analysis<br>Population/Dataset |
|---|---|---|
| 1621 5 | Subject Disposition | |
| 10.2.1 – 3 | Subject Dispositions | All Subjects |
| | Withdrawals | All Subjects |
| 1622-I | nclusion and Exclusion Criteria | |
| 10.2.2 | Inclusion and Exclusion Criteria | All Subjects |
| 16.2.3 – I | Demography and Baseline Characteristics | |
| | Demography and Baseline Characteristics | All Subjects |
| 16.2.4 – N | Medical History and medications | |
| | Medical history and Complications | All Subjects |
| | Allergic History | All Subjects |
| | Prior and Concomitant Medications | All Subjects |
| 16.2.5 – I | Exposure and Compliance | |
| | Study Drug Exposure and Compliance | All Subjects |
| 16.2.6 – I | Pharmacokinetics | |
| | List of Blood Collection Time for Pharmacokinetic Evaluation | All Subjects |
| | List of Plasma Concentrations | All Subjects |
| | List of Plasma Pharmacokinetic Parameters | All Subjects |
| | List of Ctrough Ratio | All Subjects |
| 16.2.7 – 1 | Adverse Events | |
| | Adverse Events | All Subjects |
| 16.2.8 – I | Laboratory Parameters | |
| | Laboratory Tests - Haematology | All Subjects |
| | Laboratory Tests - Biochemistry | All Subjects |
| | Laboratory Tests - Coagulation | All Subjects |
| | Laboratory Tests - Urinalysis | All Subjects |
| 16.2.9 – 0 | Other safety assessments | |
| | Physical Examinations, Weight and BMI | All Subjects |
| , | Vital Signs | All Subjects |
| | 12-Lead ECG | All Subjects |
| | Sensory Tests | All Subjects |

#### 12.2 Tables

| No. | Title of table | Analysis Population/Dataset |
|---|---|---|
| 14.1 – Stu | dy | |
| • | Subjects Dispositions and Analysis Population | All Subjects |
| | Demography and Baseline Characteristics | Safety |
| - | Summary of Prior Medications | Safety |
| | Summary of Concomitant Medications | Safety |
| 14.2 – Pha | rmacokinetics | |
| | Descriptive Statistics for Plasma Concentrations | PK |
| _ <del></del> | Descriptive Statistics for Plasma Pharmacokinetic Parameters | PK |
| | Dose proportionality in Pharmacokinetics using the power model | PK |
| | Evaluation of food effect by plasma pharmacokinetic parameters | PK |
| | Evaluation of racial differences by Plasma Pharmacokinetic parameters | PK |
| | Evaluation of difference by adding thickener by Plasma<br>Pharmacokinetic parameters | PK |
| | Descriptive Statistics for Ctrough Ratio | PK |
| | Evaluation of Linearity | PK |
| | Evaluation of Accumulation | РК |
| 14.3 – Saf | | |
| | Summary of Treatment Emergent Adverse Events | Safety |
| | Incidence and Frequency of Treatment Emergent Adverse | Safety |
| | Events by System Organ Class and Preferred Term | |
| | Incidence and Frequency of Treatment Emergent Adverse<br>Events by System Organ Class, Preferred Term and<br>Severity | Safety |
| | Incidence and Frequency of Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Relation to Study Drug | Safety |
| | Summary of Laboratory Tests - Haematology | Safety |
| | Summary of Laboratory Tests - Biochemistry | Safety |
| | Summary of Laboratory Tests - Coagulation | Safety |
| | Summary of Laboratory Tests - Urinalysis | Safety |
| | Shift table of Laboratory Tests - Urinalysis | Safety |
| | Weight | Safety |
| | Vital Signs | Safety |
| | 12-Lead ECG | Safety |
| | Summary of Sensory Tests - Vibratory Sensation | Safety |
| | Shift table of Sensory Tests - Numbness and Staggering | Safety |
| | Frequency of Abnormal values in Sensory Tests - Numbness and Staggering | Safety |

#### 12.3 Figures

| No. | Title of figure | Notes |
|---|---|---|
| SALESCON AND ACCUMENTS OF ACT | macokinetics | |
| | Profile of Mean Plasma Concentrations | PK |
| | Scatter plot of C <sub>max</sub> , AUC <sub>0-Sh</sub> , AUC <sub>0-last</sub> and | PK |
| | AUC <sub>0-∞</sub> vs dose | |
| | Box and Whisker Plot of C <sub>max</sub> /D, AUC <sub>0-8h</sub> /D, | PK |
| | AUC <sub>0-last</sub> /D and AUC <sub>0-∞</sub> /D by Dose | |
| | Box and Whisker Plot of Cmax, AUC0-last and | PK |
| | AUC <sub>0∞</sub> by Fasted and Fed Administration | |
| | Forest Plot of Ratio of Geometric LSmeans | PK |
| 1 | between Fasted and Fed Administration for | |
| | C <sub>max</sub> , AUC <sub>0-last</sub> and AUC <sub>0-∞</sub> | |
| | Box and whisker plot of C <sub>max</sub> *kg, AUC <sub>0-last</sub> *kg | PK |
| | and AUC <sub>0-∞</sub> *kg by Racial Differences | |
| | Box and whisker plot of Cmax, AUColast and | PK |
| | AUC <sub>0∞</sub> by Racial Differences | |
| | Box and whisker plot of C <sub>max</sub> , AUC <sub>0-last</sub> and | PK |
| | AUC <sub>0-∞</sub> by Presence or Absence | |
| | Profile of Ctrough | PK |
| | Forest Plot of Linearity Factor | PK |
| | Forest Plot of Ratio of Accumulation | PK |
| 16.2.6 – Pl | narmacokinetics | |
| | Profile of Individual Subject Plasma | PK |
| | Concentrations | |

#### 13. REVISION HISTORY FOR SAP AMENDMENTS

Version 2.0 (9 October, 2018)

It reflected the results of the data review meeting on

In APPROVAL FORM, the change of the person in charge of MTPC Statistics Reviewer was reflected.

In Section 7.7.8 and Section 7.7.9, the two-sided confidence level of the confidence interval has been changed from 90% to 95%.

In Section 7.8.1, the method to calculate the duration of the AE and the time from start of the IMP to AE occurrence has been changed from date to date/time.

#### APPENDIX 1 – PHARMACOKINETIC PARAMETER CALCULATIONS

- Actual blood sampling times for the assay of edaravone will be used in the calculation of pharmacokinetic parameters

Protocol No. MT-1186-J01

Date: 9 October, 2018

- All concentrations below the LLOQ will be set at zero for pharmacokinetic calculations
- When  $\lambda_z$  is missing (or cannot be determined), AUC<sub>0- $\infty$ </sub>, AUC%<sub>ex</sub>, MRT<sub>0- $\infty$ </sub>, CL/F, V<sub>ss</sub>/F, V<sub>z</sub>/F, Lower limited of  $\lambda_z$ , Upper limited of  $\lambda_z$  and Number of  $\lambda_z$  points will not be calculated

| Parameters | Unit | Calculation | Part 1 | Part 2 |
|---|---|---|---|---|
| AUC <sub>0-last</sub> | h•ng/mL | will be calculated using the linear trapezoidal method and actual times | | |
| AUC <sub>0-last</sub> /D<br>AUC <sub>0-last</sub> *kg | h•ng/mL/mg<br>h•ng/mL•kg | $AUC_{0-last} = \sum_{i=1}^{n} \frac{t_i - t_{i-1}}{2} (C_{i-1} + C_i)$ | * | <u>-</u> |
| | | /D: Divided by daily doses *kg: Multiplied by body weight on Day -1 | | |
| AUC <sub>0-8h</sub> | h•ng/mL | will be calculated using time until 8h drug concentration. | | |
| AUC <sub>0-8b</sub> /D | h•ng/mL/mg | /D: Divided by daily doses | * # | - |
| AUC <sub>0-8h</sub> *kg | h•ng/mL•kg | *kg: Multiplied by body weight on Day -1 | i | |
| AUC <sub>0-12h</sub><br>AUC <sub>0-24h</sub> | h•ng/mL | will be calculated using time until 12 or 24h drug concentration. | * . | * |
| AUC <sub>0-∞</sub> /D<br>AUC <sub>0-∞</sub> *kg | h•ng/mL<br>h•ng/mL/mg<br>h•ng/mL•kg | $AUC_{0-\infty} = AUC_{0-last} + \frac{C_{last}}{\lambda_z}$ /D: Divided by daily doses | * | * |
| AUC <sub>0-τ</sub> | h•ng/mL | *kg: Multiplied by body weight on Day -1 will be calculated using time until last quantifiable drug concentration. | - | * |
| AUC% <sub>ex</sub> | % | $AUC\%_{ex} = \frac{AUC_{0-\infty} - AUC_{0-last}}{AUC_{0-\infty}} \times 100$ | * | * |
| C <sub>max</sub> /D<br>C <sub>max</sub> *kg | ng/mL<br>ng/mL/mg<br>ng/mL•kg | will be determined using maximum drug concentration /D: Divided by daily doses *kg: Multiplied by body weight on Day -1 | * | * |
| Ctrough,DayX Ctrough,ss | ng/mL | will be determined using minimum drug concentration by each dosing day X: Each dosing day after first dose (pre-dose on Day 2 to 5) ss: After dosing interval time on last dosing day (24h on Day 5) | - | * |

| Parameters | Unit | Calculation | Part 1 | Part 2 |
|---|---|---|---|---|
| CL/F | L/h | will be calculated for unchanged edaravone only | | |
| | | Dose | * | - |
| | | $CL/F = \frac{Dose}{AUC_{0-\infty}}$ | | |
| CT /E | L/h | will be calculated for unchanged edaravone only | | |
| CL <sub>ss</sub> /F | L/II | | _ | * |
| | | $CL_{ss}/F = \frac{Dose \text{ (single dose)}}{AUC_{0-\tau}}$ | | |
| | | AUC <sub>0-τ</sub> | | |
| $\lambda_z$ | /h | The exponential rate constant of the terminal phase, $\lambda_z$ , | • | |
| | | will be estimated by log-linear regression, if determinable. | | |
| | | The number of data points included in the regression will be determined by visual inspection. Wherever possible, a | | |
| | | minimum of 3 data points will be used in the estimation of | <u> </u> | |
| | | $\lambda_{\mathbf{z}}$ . | | |
| | | During the analysis, this calculation method repeats regressions using the last three points with non-zero | | |
| | | concentrations, then the last four points, last five, etc. | | |
| | | Points prior to C <sub>max</sub> or prior to the end of infusion will not | | |
| | | be used unless the user specifically requests that time | | |
| | | range. Points with a value of zero for the dependent | * | * |
| | | variable will be excluded. For each regression, an adjusted R <sup>2</sup> will be computed | | |
| | | Adjusted $R^2 = 1 - \frac{(1 - R^2) + (n - 1)}{(n - 2)}$ | | |
| | | where n is the number of data points in the regression and | | |
| | | $\mathbb{R}^2$ is the square of the correlation coefficient. | | |
| | | The regression with the largest adjusted R <sup>2</sup> will be | | - |
| | | selected to estimate $\lambda z$ , with these caveats: | | |
| | | If the adjusted R <sup>2</sup> does not improve, but is within 0.0001 | | |
| | | of the largest adjusted R <sup>2</sup> value, the regression with the | | |
| | | larger number of points will be used. $\lambda_z$ must be positive, | | |
| | | and calculated from at least three data points. | · | <u> </u> |
| Lower | h | will be determined using lower limit on time to be | * | * |
| limited of $\lambda_z$ | | included in the calculation of $\lambda_z$ | | |
| LF | - | AUC. (last dose) | | |
| | | $LF = \frac{AUC_{0-\tau} \text{ (last dose)}}{AUC_{0-\infty} \text{ (first dose)}}$ | _ | * |
| | | | - | |
| | | τ : Dosing interval | | |
| MRT <sub>0-∞</sub> | h | will be calculated for unchanged edaravone only | | |
| 1411(1.0.00 | •• | n | | |
| | | $AUMC_{0-\infty} = \sum_{i=1}^{n} \frac{(t_i - t_{i-1})(t_i \times C_i + t_{i-1} \times C_{i-1})}{2}$ | | |
| | | $+\frac{t \times C_t}{\lambda_z} + \frac{C_t}{(\lambda_z)^2}$ | * | - |
| | | $\lambda_z (\lambda_z)^2$ | | |
| | | } | | |
| | | $MRT_{0-\infty} = \frac{AUMC_{0-\infty}}{AUC_{0-\infty}}$ | | |
| | | AUC <sub>0-∞</sub> | | |
| MRT <sub>ss</sub> | h | 911 1 1 1 1 6 | | * |
| | | will be calculated for unchanged edaravone only | 1 | " |

| | | PK Parameter Calculations | | 1000 |
|---|---|---|---|---|
| Parameters | Unit | Calculation | Part 1 | Part 2 |
| | | $\begin{aligned} \text{AUMC}_{0-\tau} &= \sum_{i=1}^{n} \frac{(t_i - t_{i-1})(t_i \times C_i + t_{i-1} \times C_{i-1})}{2} \\ \text{MRT}_{ss} &= \frac{\text{AUMC}_{0-\tau} + \tau \times (\text{AUC}_{0-\infty} - \text{AUC}_{0-\tau})}{\text{AUC}_{0-\tau}} \end{aligned}$ | · | |
| Number of $\lambda_z$ points | - | will be determined using number of points used in computing $\lambda_z$ . If $\lambda_z$ cannot be estimated, zero. | * | * |
| RA | - | $RA = \frac{AUC_{0-\tau} \text{ (last dose)}}{AUC_{0-\tau} \text{ (first dose)}}$ | - | * |
| | | τ : Dosing interval | | |
| t <sub>1/2</sub> | h | $t_{1/2}$ will be determined as: $t_{1/2} = \frac{\log_e(2)}{\lambda_z}$ | * | * |
| t <sub>max</sub> | h | will be determined using time to maximum drug concentration | * | * |
| Upper limited of λ <sub>z</sub> | h | will be determined using upper limit on time to be included in the calculation of $\lambda_{\mathbf{z}}$ | * | * |
| V <sub>ss</sub> /F | L | will be calculated for unchanged edaravone only $V_{ss}/F = MRT_{ss} \times CL_{ss}/F \label{eq:vss}$ | - | * |
| V <sub>z</sub> /F | L | will be calculated for unchanged edaravone only $V_z/F = CL/F \times \frac{1}{\lambda_z}$ | * | - |



### Statistical Analysis Plan for ECGs

Mitsubishi Tanabe Pharma Corporation

Phase I Study of Oral Edaravone in Healthy Adult Males (Single- and Multiple-Dose Study)

Protocol ID: MT-1186-J01

Author , MD

Date of Issue: 26 July 2018

NCT number: NCT04481750






| • | | | • | | 1 1 |
|---|-----|------------|-----|-----|-----|
| | 1 | CT. | Λŧ | Ta | n |
| | 4 . | <b>31.</b> | .,, | - 4 | |

| Table 3: Goodness of Fit Plots | 15 |
|---|---|
| Table 4: ECG Evaluable Population | 17 |
| Table 5: Summary Statistics for QTcF and Change of QTcF from Baseline | e (msec) 18 |
| Table 6: Summary Statistics for HR and Change of HR from Baseline (bp | m)20 |
| Table 7: Summary Statistics for PR and Change of PR from Baseline (mse | ec) 20 |
| Table 8: Summary Statistics for QRS and Change of QRS from Baseline ( | (msec) 20 |
| Table 9: Edaravone QTcF Regression Analysis: Estimated Mean Place | bo-adjusted Change of |
| QTcF from Baseline at Various Edaravone Concentration Levels and 2 | -sided 90% Confidence |
| Bounds (msec) | 21 |
| Table 10: Edaravone HR Regression Analysis: Estimated Mean Placebo- | adjusted Change of HR |
| from Baseline at Various Edaravone Concentration Levels and 2-sided 9 | 0% Confidence Bounds |
| (msec) | 22 |
| Table 11: Edaravone PR Regression Analysis: Estimated Mean Placebo- | adjusted Change of PR |
| from Baseline at Various Edaravone Concentration Levels and 2-sided 9 | 0% Confidence Bounds |
| (msec) | 22 |
| Table 12: Edaravone QRS Regression Analysis: Estimated Mean Place | ebo-adjusted Change of |
| QRS from Baseline at Various Edaravone Concentration Levels and 2 | -sided 90% Confidence |
| | 22 |
| Table 13: Edaravone QTcF Regression Analysis: Regression Statistics | 23 |
| Table 14: Edaravone HR Regression Analysis: Regression Statistics | 23 |
| Table 15: Edaravone PR Regression Analysis: Regression Statistics | 23 |
| Table 16: Edaravone QRS Regression Analysis: Regression Statistics | 23 |
| Table 17: LS Mean Changes from Baseline in QTcF for Edaravone and | l Placebo and LS Mean |
| Placebo-subtracted Changes from Baseline in QTcF and 1-sided 95% Up | |
| (msec) | |
| Table 18: LS Mean Changes from Baseline for HR for Edaravone and | |
| Placebo-subtracted Changes from Baseline in QTcF and 2-sided 90% Co. | nfidence Bounds (msec) |
| 1 idees Stoffdeted Changes from Baseman in \$2.51 and 2 states \$7.5 and | |
| Table 19: LS Mean Changes from Baseline for PR for Edaravone and | |
| Placebo-subtracted Changes from Baseline in QTcF and 2-sided 90% Co | nfidence Bounds (msec) |
| Theodor subtracted changes from Substitute in \$2.50 miles 2.50 miles | |
| Table 20: LS Mean Changes from Baseline for QRS for Edaravone and | d Placebo and LS Mean |
| Placebo-subtracted Changes from Baseline in QTcF and 2-sided 90% Up | oper Confidence Bounds |
| (msec) | |
| Table 21: Number (%) of Subjects with a QTcF Interval >450 msec | |
| Table 22: Number (%) of Subjects with a QTcF Interval >480 | 27 |
| Table 23: Number (%) of Subjects with a QTcF Interval >500 msec | 27 |
| Table 24: Number (%) of Subjects with a QTcF Interval Change from | Baseline in OTcF >30 |
| Table 24. Number (70) of Subjects with a Q1er interval change from | 2.7 |
| msec | from Baseline in OTcF |
| >60 msec | 27 |
| Table 26: Number (%) of Subjects with HR <40 bpm after a decrease | e of HR >20 hom from |
| Reseline | 27 or the <u>2</u> 20 opin from 27 |

| Table 27: Number (%) of Subjects with HR >110 bpm after an increase of HR ≥20 bpm from Baseline |
|---|
| Table 28: Number (%) of Subjects with PR interval of <100 msec after a decrease of PR interval ≥25% from Baseline |
| Table 29: Number (%) of Subjects with PR interval of >220 msec after an increase of PR interval |
| ≥25% from Baseline |
| Table 30: Number (%) of Subjects with QRS duration >120 msec after an increase of QRS |
| duration ≥25% from Baseline |
| Table 31: Subjects with an ECG Diagnostic Finding Not Present at Baseline Tracings |
| List of Figures |
| Figure 1: Study Flow Chart9 |
| Figure 2: Arithmetic Mean QTcF (msec) |
| Figure 3: Arithmetic Mean HR (bpm) |
| Figure 4: Arithmetic Mean PR (msec) |
| Figure 5: Arithmetic Mean QRS (msec) |
| Figure 6: Arithmetic Mean Change from Baseline in QTcF |
| Figure 7: Arithmetic Mean Change from Baseline in HR (bpm) |
| Figure 8: Arithmetic Mean Change from Baseline in PR (msec) |
| Figure 9: Arithmetic Mean Change from Baseline in QRS (msec) |
| Figure 10: Edaravone QTcF-Concentration Regression Analysis: Change of QTcF from Baseline |
| versus Edaravone Concentration, Combined Doses: Slope (if linear) and 2-sided 90% |
| Confidence Bounds of the Slope (msec) |
| Figure 11: Edaravone HR-Concentration Regression Analysis: Change of QTcF from Baseline |
| versus Edaravone Concentration, Combined Doses: Slope (if linear) and 2-sided 90% |
| Confidence Bounds of the Slope (msec) |
| Figure 12: Edaravone PR-Concentration Regression Analysis: Change of QTcF from Baseline |
| versus Edaravone Concentration, Combined Doses: Slope (if linear) and 2-sided 90% |
| Confidence Bounds of the Slope (msec) |
| Figure 13: Edaravone QRS-Concentration Regression Analysis: Change of QTcF from Baseline |
| versus Edaravone Concentration, Combined Doses: Slope (if linear) and 2-sided 90% |
| Confidence Bounds of the Slope (msec) |
| Figure 14: Edaravone QTcF-Concentration Regression Analysis: From Slope and 2-sided 90% |
| Confidence Bounds of the Slope (if linear), Combined Doses: Estimated Mean Placebo-adjusted |
| Change of QTcF from Baseline at Geometric Mean Cmax Edaravone Concentration Levels and 2-sided 90% Confidence Bounds (msec) |
| 2-sided 90% Confidence Bounds (msec) |
| 90% Confidence Bounds of the Slope, Combined Doses: Estimated Mean Placebo-adjusted |
| Change of QTcF from Baseline at Geometric Mean Cmax Edaravone Concentration Levels and |
| 2-sided 90% Confidence Bounds (msec) |
| Figure 16: Edaravone PR-Concentration Regression Analysis: From Slope (if linear) and 2-sided |
| 90% Confidence Bounds of the Slope, Combined Doses: Estimated Mean Placebo-adjusted |
| Change of QTcF from Baseline at Geometric Mean Cmax Edaravone Concentration Levels and |
| 2-sided 90% Confidence Bounds (msec) |

| Figure 17: Edaravone QRS-Concentration Regression Analysis: From Slope (if linear) and 2-sided 90% Confidence Bounds of the Slope, Combined Doses: Estimated Mean Placebo-adjusted Change of QTcF from Baseline at Geometric Mean Cmax Edaravone Concentration Levels and 2-sided 90% Confidence Bounds (msec) |
|---|
| Figure 18: Change of HR from Baseline versus Edaravone Concentration and 2-sided 90% |
| Confidence Bounds of the Slope (msec) |
| Figure 19: QTcF vs. RR and 2-sided 90% Confidence Bounds of the Slope (msec) |
| Figure 20: Hysteresis Analysis: Highest Edaravone Dose Group: LS Mean Placebo-adjusted |
| Change from Baseline (ΔΔQTcF) (msec) and Edaravone Concentration (ng/mL) |
| Figure 21: Paired ΔQTc and Concentration with Loess Smooth Line and 95% Confidence |
| Intervals and Linear Regression |
| Figure 22: Paired $\Delta$ HR and Concentration with Loess Smooth Line and 95% Confidence |
| Intervals and Linear Regression |
| Figure 23: Paired APR and Concentration with Loess Smooth Line and 95% Confidence |
| Intervals and Linear Regression |
| Intervals and Linear Regression |
| Intervals and Linear Regression |
| Figure 25: Edaravone QTcF-Concentration Regression Analysis: Model Predicted vs Observed |
| AOTcF |
| Figure 26: Edaravone HR-Concentration Regression Analysis: Model Predicted vs Observed |
| $\Delta QHR$ 39 |
| Figure 27: Edarayone PR-Concentration Regression Analysis: Model Predicted vs Observed |
| ΔPR |
| Figure 28: Edaravone QRS-Concentration Regression Analysis: Model Predicted vs Observed |
| $\Delta QRS$ |
| ΔQRS |
| Residuals 39 |
| Figure 30: Edaravone HR-Concentration Regression Analysis: Quantile-Quantile Plot of Residuals |
| 10014440 |
| Figure 31: Edaravone PR-Concentration Regression Analysis: Quantile-Quantile Plot of |
| Residuals Concentration |
| Figure 32: Edaravone QRS-Concentration Regression Analysis: Quantile-Quantile Plot of |
| Residuals |
| Figure 34: Edaravone HR-Concentration Regression Analysis: Concentration vs Residuals 39 |
| Figure 35: Edaravone PR-Concentration Regression Analysis: Concentration vs Residuals 39 |
| Figure 36: Edaravone QRS-Concentration Regression Analysis: Concentration vs Residuals 39 |
| Figure 37: Edaravone QTcF Regression Analysis: Baseline QTcF vs Residuals |
| Figure 38: Edaravone HR Regression Analysis: Baseline HR vs Residuals |
| Figure 39: Edaravone PR Regression Analysis: Baseline PR vs Residuals |
| Figure 40: Edaravone QRS Regression Analysis: Baseline QRS vs Residuals Residuals |
| Figure 41: Edaravone QTcF Regression Analysis: Active Treatment vs Residuals |
| Figure 42: Edaravone HR Regression Analysis: Active Treatment vs Residuals |
| Figure 43: Edaravone PR Regression Analysis: Active Treatment vs Residuals |

| igure 44: Edaravone QRS Regression Analysis: Active Treatment vs Residuals | 39 |
|---|---|
| gure 45: LS Mean Placebo-adjusted Change from Baseline in QTcF and 1-sided Upper 95 | 5% |
| Confidence Bounds (msec) | |
| Figure 46: LS Mean Placebo-adjusted Change from Baseline in HR and 2-sided 90% C | |
| Confidence Bounds (bpm) | |
| Figure 47: LS Mean Placebo-adjusted Change from Baseline in PR and 2-sided 90% C | CIs |
| Confidence Bounds (msec) | |
| figure 48: LS Mean Placebo-adjusted Change from Baseline in QRS and 2-sided 90% C | |
| Confidence Bounds (msec) | 40 |
| List of Appendices | |
| Appendix 1: Listing of Individual Subject ECG Data | 41 |
| Appendix 2: Listing of Individual Subject Change of ECG Intervals (Δ) and Edaravo | ne |
| Concentration | |
| Appendix 3: Listing of Abnormal ECG Morphologies | 43 |






MITSUBISHI TANABE PHARMA CORPORATION CONFIDENTIAL



Edaravone, a free radical scavenger, has been approved as for the treatment of amyotrophic lateral sclerosis.

Nevertheless, IV infusion places a large burden on patients with ALS; therefore, there is a need for more convenient oral agents. An oral formulation of edaravone is to be developed and MT-1186-J01 is the first study to assess bioavailability in humans.

This protocol will assess the effects of single or multiple dose of edaravone or placebo given orally and will assess the pharmacodynamics of edaravone versus placebo on the QT interval of the electrocardiogram (ECG) corrected for heart rate (HR) by Fridericia's formula (QTcF) in healthy adult subjects, to meet the objectives of a formal QT/QTc study, as required in accordance with ICH E14<sup>1</sup>. The study is designed to comply with the ICH E14 guidance, specifically the update of June 2017<sup>2</sup>, in utilizing exposure-response analysis as the method for primary analysis.

This document outlines the planned analysis of the pharmacodynamic (PD) ECG data.

### 2. STUDY DESIGN

This is a Phase 1, placebo-controlled, randomized, single-blinded study of the effect of single and multiple doses of edaravone versus placebo on the ECG in healthy adult male volunteers. This study will be performed using a placebo-controlled, randomized, single-blind design, and consists of Part 1 (single-dose study) and Part 2 (multiple-dose study).

Pharmacodynamic determinations will be based on the concentration of unchanged edaravone. While the concentrations of the major metabolites, sulfate conjugate and glucuronide conjugate, will be measured, as stated in the protocol, these are not consider active metabolites, as "neither a free radical scavenging effect nor a lipid peroxidation inhibitory effect have been observed".

The flow of planned cohort transition in this study is shown in Figure 1. Except in Cohorts S3-1 and S3-2, no subjects are planned to receive study drug in multiple cohorts.

<sup>2</sup> ICH HARMONISED TRIPARTITE GUIDELINE:— E14. Update R3: June 2017.

<sup>&</sup>lt;sup>1</sup> International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use - ICH HARMONISED TRIPARTITE GUIDELINE: The Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs – E14. 12 May 2005.



<u>53-2</u> 800 mg\* Single dose (after meal) <u>\$4</u> S3-1 **S1** 240 mg\* Single dose (fasting) 1600 mg\* Singe dos (fasting) 60 mg Single dos (fasting) 800 mg\* Single dose (fasting) apanese P=6:2 Japanese E:P=6:2 <u>S7</u> 800 mg\* Single dose (fasting) White 2400 mg\* Multiple dose Cohort No., Dose /day. (fasting /after meal), race, randomization rate. (E:edaravone, P:Placebo) Temporary dose. Dose will be decided based on PK and safety data in the previous cohort.

Figure 1: Study Flow Chart

### **2.1. Doses**

The actual doses to be administered to each cohort are as follows:

Dose, Dosing Regimen, and Duration (Single-dose study [Part 1])

| Cohort | Dose | Condition of | Race | Duration | No. of subjects | |
|---|---|---|---|---|---|---|
| | | administration | | | Edaravone | Placebo |
| S1 | 60 mg | | | 1 day | 6 | 2 |
| S2 | 120 mg | Fasting | | 1 day | 6 | 2 |
| S3-1 | 200 | | lananasa | 1 day | 6 | 2 |
| S3-2 | 200 mg | After a meal | Japanese | 1 day | 0 | |
| S4 | 300 mg | | | 1 day | 6 | 2 |
| S5 | 300 mg | Fasting | , | 1 day | 6 | 2 |
| S6 | 30 mg | | | 1 day | 6 | 2 |
| S7 | 200 mg | | Caucasian | 1 day | 6 | 2 |

# Dosing Regimen, and Duration (Multiple-dose study [Part 2])

| Cohort | Dose | Frequency of | Duration | No. of subjects | |
|---|---|---|---|---|---|
| | | administration | | Edaravone | Placebo |
| M1 | 120mg | Once daily | 5 days | 6 | 3 |
| M2 | 200 mg | Once daily) | 5 days | 6 | 3 |

### 2.2. Subjects

The study will enrol 74 subjects.

• Part 1 (single-dose study): 56 subjects (8 subjects per cohort: 6 subjects in the edaravone group and 2 subjects in the placebo group)



• Part 2 (multiple-dose study): 18 subjects (9 subjects per cohort: 6 subjects in the edaravone group and 3 subjects in the placebo group)

### 2.3. Objective

To evaluate QTcF prolongation and proarrhythmic potential for edaravone.

### 2.4. Pharmacodynamic Endpoints

Analysis of ECGs for pharmacodynamic (PD) endpoints will be limited to Part 1 Japanese Cohorts given single doses, fasting, in cohorts S4, S5 and S6. Total subjects in the PD population will be 24: 18 active and 6 placebo.

ECG parameters studied will be HR, QTcF, PR interval (PR) and QRS duration (QRS).

### 2.5. PD ECG and PK SCHEDULE

In Part 1, continuous 12-lead Holter data will be obtained for Cohorts S4, S5, and S6 on Day 1 from at least 1 hour predose to 48 hours postdose. PD ECGs will be extracted from the Holter data at multiple timepoints after dosing and centrally read by the ECG Core Laboratory, with results available after the completion of the study. A single cardiologist will be assigned to read all ECGs from any individual subject, blinded to treatment and timepoint sequence. Intervals will be determined in a semi-automated fashion using a superimposed global 12-lead display of the median beats from each lead.

On Day 1, Baseline ECGs will be extracted in triplicate during three 5-minute observation periods starting at 45, 30 and 15 minutes prior to oral dosing; and during each 5-minute observation periods starting at 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36 and 48 hours after the start of oral dosing on Day 1.

Blood samples will be collected on Day 1 pre-dose and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36 and 48 hours post-dose.

For the purpose of maintaining the blind, blood PK samples will be collected from all subjects, but only PK samples from the edaravone dose groups will be analyzed for edaravone.

### 3. ANALYSIS VARIABLES

All ECG interval data will represent the means of up to three individual tracings, based on ECGs extracted from the Holter data approximately one minute apart. The formula to be used for all analyses of corrected QT data is:

Fridericia correction:  $QTcF = QT/RR^{(1/3)}$  (assumes RR to be in units of seconds).

Within a set of triplicate ECG measurements at each time point, each individual QT and RR will be used to calculate a QTcF interval. These individual QTcF intervals across the triplicates will then be averaged for analysis.



ECG morphologies will be assessed based on each of the triplicate ECGs separately at each timepoint.

### 4. ANALYSIS POPULATIONS

The definitions of the analysis sets are provided below.

- Safety analysis set
  The safety analysis set will consist of all subjects who received at least 1 dose of the study
  drug.
- PK analysis set The PK analysis set will consist of all subjects who received at least 1 dose of the study drug and had evaluable PK data.
- PD analysis set
  The PD analysis set will consist of all subjects who received at least 1 dose of the study drug
  and had evaluable PD data.

Any determination of subjects to be excluded will be at the direction of the sponsor, prior to the database lock.

### 5. Assessment of ECGs

### 5.1. ECG Assessment

### 5.1.1. Primary Assessment

For Cohorts S4, S5, and S6:

The primary outcome is to determine cardiac repolarization effects is the relationship of change from Baseline in QTcF with placebo adjustment ( $\Delta\Delta$ QTcF) and concentration of edaravone.

### 5.1.2. Secondary Assessments by Timepoint and by Treatment

For Cohorts S4, S5, and S6:

- Assessment of mean QTcF, and mean changes from Baseline in QTcF ( $\Delta$ QTcF), and LS mean  $\Delta\Delta$ QTcF
- Relationship of change from Baseline in HR, PR and QRS with placebo adjustment and concentration of edaravone.
- Assessment of mean HR, PR and QRS, and mean changes from Baseline, and LS mean placebo-adjusted changes.
- Proportion of subjects with a QTcF interval ≥450, ≥480, and ≥500 msec
- Proportion of subjects with an increase from Baseline in QTcF interval of >30 and
   >60 msec
- Proportion of subjects with HR, PR interval, or QRS duration abnormalities (based on the Core ECG Laboratory's standard clinically relevant values and clinically relevant changes):




- o HR <40 bpm after a decrease of HR ≥20 bpm from Baseline, or HR >110 bpm after an increase of HR ≥20 bpm from Baseline
- o PR interval of <100 msec after a decrease of PR interval ≥25% from Baseline, or PR interval of >220 msec after an increase of PR interval ≥25% from Baseline
- o Change of QRS duration ≥25% from Baseline reaching a QRS ≥120 msec
- Proportion of subjects with an emergent ECG diagnostic abnormality

### 6. STATISTICAL METHODS

All values will represent means of triplicate ECGs at each timepoint. The statistical analysis will be performed using SAS® Version 9.2 or higher. The PD analysis set will be used for all definitive cardiac analysis. Edaravone concentration assessments for the PK analysis set will be combined with the PD ECG values for the PD analysis set. Unless stated otherwise, all formal statistical tests will be done at the 5% two-sided significance level. Point estimates will have 2-sided 95% confidence intervals (CIs).

### 6.1. Pooled ECG Data

Data for ECG intervals for the placebo dose groups will each be combined from subjects in all three cohorts.

### 6.2. Baseline

Based on all of the ECG interval values for each subject collected prior to dosing (up to 9, i.e., three timepoints with triplicate ECGs at each) subject-specific baseline the mean of the interval values will be calculated for each parameter. The subject-specific Baseline diagnostic findings will include each abnormality found on any of the predose ECGs for that subject.

### 6.3. Interval Summary Statistics

Interval analyses by timepoints will be presented in summary statistics (number (N), mean, median, minimum (min), maximum (max), standard deviation [SD], 2-sided 90% CI range for HR, PR interval, QRS duration, and QTcF intervals in tables and displayed in figures by treatment for the: (1) absolute values at Baseline and for each day by timepoint; and (2) change from Baseline for each day by timepoint.

### 6.4. OTcF-Concentration Regression Analysis

The primary outcome endpoint will be based on an analysis of the regression relationship between  $\Delta QTcF$  and the concentration of edaravone at matching times post-dose, including adjustment for placebo subjects, to provide estimates equivalent to  $\Delta\Delta QTcF$ , as follows:

- All paired values of ΔQTcF and concentration, from all subjects and timepoints (hours), will be included (edaravone and placebo-treated subjects) with concentration values of lower than lower limit of quantification and placebo concentration values set to 0
- A linear mixed effects model will be performed with: (1) ΔQTcF as the dependent variable, edaravone plasma concentration and Baseline QTcF (subjects baseline overall mean baseline for all subjects) as continuous covariates; (2) time (hours), treatment (any



dose level of edaravone vs placebo) as categorical factors; and (3) a random intercept and slope per subject

- The slope of the regression relationship and the 2-sided 95% CI of the slope will be calculated.
- From PK data (separate from the model) the geometric mean (of each individual subject's values of)  $C_{max}$  of edaravone, for each dose level, will be calculated; as well as the quintiles of edaravone concentration for the three dose levels combined
- At these geometric mean  $C_{max}$  values calculated from the regression of dQTcF vs concentration (which includes a treatment effect, time effect, baseline QTcF effect, and random slope and intercept effects), point estimates for placebo-adjusted changes of QTcF from Baseline (equivalent to  $\Delta\Delta$ QTcF) and the corresponding 2-sided 90% CIs will be constructed
- If the upper bounds of the CIs at the geometric mean C<sub>max</sub> levels for edaravone are both <10 msec, then it will be concluded that the QTc interval prolongation is not clinically meaningful



### Model Information

| Data Set | WORK.TEST |
|---------------------------|---------------|
| Dependent Variable | QTcF |
| Covariance Structure | Unstructured |
| Subject Effect | Id |
| Estimation Method | REML |
| Residual Variance Method | Profile |
| Fixed Effects SE Method | Kenward-Roger |
| Degrees of Freedom Method | Kenward-Roger |

If the model fails to converge, alternate approaches will be pursued.

### 6.5. Exploration of Model

### 6.5.1. Heart Rate Effects

The model assumptions will be assessed by inspection of slope and 2-sided 90% CIs, without formal statistics, to show that:




- there is an insignificant effect of edaravone on change of HR (plot of  $\Delta$ HR vs. concentration)
- there is adequate normalization of QTcF for RR (plot of QTcF vs. RR),

### 6.5.2. Hysteresis

If the by-timepoint analysis (see below Section 6.6.1) cannot exclude an effect of  $\Delta\Delta QTcF$  <10 msec, hysteresis will be examined by simultaneously displaying in a figure the time course of mean  $\Delta\Delta QTcF$  and the concentration of edaravone for the highest dose edaravone dose group. A delay of maximum  $\Delta\Delta QTcF$  with respect to the maximum concentration of edaravone >1.0 hour will be considered an indication of hysteresis. In addition, a scatter plot of paired  $\Delta QTc$  and concentration with loess smooth line and 95% confidence intervals and linear regression line. If hysteresis is determined to be present, an alternate analysis may be explored.

### 6.5.3. Linear Model Criteria

To document the success of the *a priori* choice of linear model, a table will provide the Akaike Information Criteria (AIC) for linear, quadratic and cubic fits of the regression. If one of the alternate models provides a substantially better fit, that model will be used to derive the primary endpoint.

Per the recent recommendations<sup>3</sup>, the element shown in Table 1 will be assessed:

<sup>&</sup>lt;sup>3</sup> Garnett, C., Bonate P, et al. Scientific white paper on concentration-QTc modeling. *Journal of Pharmacokinetics and Pharmacodynamics*: https://doi.org/10.1007/s10928-017-9558-5.



**Table 1: Goodness of Fit Plots** 

| lot | Model assumption tested | What to evaluate | Model impact |
|---|---|---|---|
| Model predicted<br>versus observed<br>AQTc | Model specification is adequate. | Model and observed values should fall<br>around the line of unity without<br>evidence of systematic bias. Loess<br>smooth line with 95% CI should include<br>the unity line over range of values | Systematic bias indicates model misspecification. For example, model predictions will be negatively biased at high values when PK/PD hysteresis is ignored and model predictions will be positively biased at high values when a linear model is applied to nonlinear data |
| Quantile-Quantile plot of residuals | Residuals follow normal distribution with mean of zero | Residuals should fall on the line of unity | Heavy tails indicate model<br>misspecification. The plot does not<br>indicate source of misspecification |
| Concentrations versus residuals | Model covariates are adequate | Residuals should be randomly scattered around zero | Bias in residuals indicates model<br>misspecification. A residual plot should<br>be made for each model parameter |
| Baseline QTc versus residuals | | The 95% CI of the loess line should include zero | |
| Time versus residuals | | | |
| Active treatment versus residuals | | | |

### 6.6. Secondary Analyses

# 6.6.1. Analysis of Central Tendency for QTcF

As a secondary analysis, but without formal hypothesis testing, an intersection-union test (whether or not one-sided 95% CI Upper Bound will be lower than 10 msec at all time-points) of  $\Delta\Delta QTcF$  will be analysed using a Mixed Model for Repeated Measures (MMRM) on the PD population. The model will include treatment and scheduled visit as fixed effects, corresponding baseline-derived parameter at baseline ECG as a covariate, and treatment-by-visit and baseline-by-visit interactions. An unstructured correlation structure will be used to model the within-subject variance covariance errors. Should the unstructured correlation structure not converge, then an AR(1) correlation matrix will be used. The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom, as follows:

• From this model the least square (LS) Mean estimates and standard deviation, difference of the means between each edaravone dose group and pooled placebo, and one-sided 95% upper confidence bounds on the difference will be presented.





In addition, an identical concentration regression analysis will be performed for HR, PR interval and QRS duration, and an identical by-timepoint analysis for HR, PR interval and QRS duration, will be presented, providing 2-sided 90% CIs rather than 1-sided upper CIs.

### 6.6.3. Categorical Analysis

Categorical analyses for QTcF interval, HR, PR interval, and QRS duration, will be presented as additional secondary endpoints:

- The proportion of subjects with a QTcF interval >450, >480, and >500 msec will be presented by dose group for each day by timepoint, separately and overall
- The proportion of subjects with a change from predose Baseline in QTcF >30 and >60 msec will be presented by dose group for each day by timepoint, separately and overall
- Proportion of subjects with HR, PR interval, or QRS duration abnormalities:
  - o HR <40 bpm after a decrease of HR ≥20 bpm from Baseline, or HR >110 bpm after an increase of HR ≥20 bpm from Baseline
  - o PR interval of <100 msec after a decrease of PR interval ≥25% from Baseline, or PR interval of >220 msec after an increase of PR interval ≥25% from Baseline
  - o QRS duration >120 msec after an increase of QRS duration ≥25% from Baseline
- The proportion of subjects, over all post-dose timepoints, with an ECG diagnostic finding not present at any of the Baseline tracings for that subject, by dose group. Diagnostic entities that represent findings based solely on numerical data, e.g., Sinus Tachycardia, will not be included.

### 7. TABLES AND LISTINGS

The following indicate the tentative doses/formulations as examples for the basic structure of tables, figures and listings. Baseline interval values will represent means of all values from the multiple ECGs predose (up to 9). All postdose interval values will represent means of triplicate ECGs at each timepoint.

**Table 2: ECG Evaluable Population** 

| Dose Group | Subjects | Males<br>(N, %) | Females (N, %) | Median<br>Age<br>(yrs) | Min<br>Age<br>(yrs) | Max<br>Age<br>(yrs) |
|---|---|---|---|---|---|---|
| Edaravone 300 mg with xanthan PO | | | | | | |
| Edaravone 300 mg without xanthan PO | | | | | | |
| Edaravone 30 mg solution PO | | | | | | |
| Combined Placebo | | | | | | |
| Overall | | | | | , | |

Table 3: Summary Statistics for QTcF and Change of QTcF from Baseline (msec)


| | Tim | Treatment ( | sod | | | | | | | | Ba | | | | | | Edaravone 30 | mg solution PO | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Timepoint | | postdose) | 8 | 12 | 24 | 36 | 48 | 36 | 48 | Baseline | 0.25 | 0.5 | 1 | 1.5 | 2 | 4 | 9 | 8 | 12 | 24 | 36 | 48 | 36 | 48 |
| | | z | | | | | | | | | | | | | | | | | | | | , | | | |
| | | Mean | | | | | | | | | | | | | | | | | | | | | | | |
| Abs | | Med | | | | | | | | | | | | - | | | | | | | | | | | |
| Absolute Values | | Min | | | | | | | | | | | | | | | | | | | | | | | |
| Values | | Мах | | | | | | | | | | | | | | | | | | | | | | | |
| | | Stq | | | | | | | | | | | | | | | | | | | | | | | |
| | 2-sided | 12 %06 | range | | | | | | | | | | | | | | | | | | | | | | |
| | | z | | | | | | | | | | | | | | | | | | | | | | | |
| | | Mean | | | | | | | | | | | | | | | | ; | | | | | | | |
| Chang | | Stq | | | | | | | | - | | | | | | | | | | | | | | | |
| <b>Change From Baseline</b> | | Med | | | | | | - | | | | | | | | | | | | | | | | | |
| Base I | | Min | | | | | | | | | | | | | | | į | | | | | | | | |
| ine | | Max | | - | | | | | | | | | | | | | | | | - | | | | | |
| | 2-sided | 30% CI | range | | | | | | | | | | | | | | | | | | | | | | |

MITSUBISHI TANABE PHARMA CORPORATION CONFIDENTIAL


| | | lreatment | | | | | | 1 | | | Combined | | | | -1 | | | <u> </u> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Timepoint | (nrs | postdose) | Baseline | 0.25 | 0.5 | П | 1.5 | 2 | 4 | 9 | 8 | 12 | 24 | 36 | 48 | 36 | 48 |
| | 2 | _ | | | | | | | | | | | | | | | | |
| | | Mean | | | | | | | | | | | | | | | | |
| \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | 2 | Med | | | | | | | | | | | | | | | | - |
| Absolute Values | 2 | | | | | | | | | | | | | | | | | |
| Values | 2 | X P I | | | | | | | | | | | | | | | | |
| | <b>7</b> | | | | | | | | | | | | | | | | | |
| | 2-sided | 30% C1 | range | | | | | | | | | | | | | | | |
| | Z | Z | | | | | | | | - | - | | | | | | | |
| | Moon | ול<br>המ | | | | | | | | | | | | | | | | |
| Chang | 7 | ם<br>ק | | | | | | | | | | | | | | | | |
| Change From Baseline | NoM | | | | | | | | | - | | | | | | | | |
| Basel 1 | Δin | | | | | | | | | | | | | | | | - | |
| ine | . N | Max | | | | | | | | | | | | | | | | |
| | 2-sided | 20.0c | range | | | | | | | | | | | | | | | |

Repeat as:

Table 4: Summary Statistics for HR and Change of HR from Baseline (bpm)
Table 5: Summary Statistics for PR and Change of PR from Baseline (msec)
Table 6: Summary Statistics for QRS and Change of QRS from Baseline (msec)


Table 7: Edaravone QTcF Regression Analysis: Estimated Mean Placebo-adjusted Change of QTcF from Baseline at Various Edaravone Concentration Levels and 2-sided 90% Confidence Bounds (msec)

| Concentration Level tration (ng/mL) By Quintiles of Concentration for All Doses Minimum 1st Quintile 2nd Quintile | (mL) | ֡֡֝֡֜֜֜֜֜֜֜֜֜֓֓֓֜֜֜֜֜֜֓֓֓֓֓֜֜֜֜֜֜֜֜֜֜֓֓֓֓֜֜֜֜ | ;<br>; | ב<br>ב<br>ב<br>ב<br>ב |
|---|---|---|---|---|
| By Quintiles of Concentration for All Doses Minimum 1st Quintile 2nd Quintile | | (msec) | 90 % CB<br>(msec) | 90 % CB (msec) |
| | | : | | |
| Minimum<br>1st Quintile<br>2nd Quintile | | | | |
| 1st Quintile<br>2nd Quintile | | | | |
| 2nd Quintile | | | | |
| 3rd Quintile | | | | |
| 4th Quintile | | | | |
| Maximum | | | | |
| By Geo. Mean of Individual Subjects' Maximum Observed | aximum ( | Observed | | |
| Plasma Concentration | | | | |
| Cmax edaravone 300 mg with | | | | |
| xanthan PO | | ; | | |
| Cmax edaravone 300 mg | | | | |
| without xanthan PO | | | | |
| Cmax edaravone 30 mg | | | | |
| solution PO | | | | |

Repeat as:

Table 10: Edaravone QRS Regression Analysis: Estimated Mean Placebo-adjusted Change of QRS from Baseline Table 8: Edaravone HR Regression Analysis: Estimated Mean Placebo-adjusted Change of HR from Baseline Table 9: Edaravone PR Regression Analysis: Estimated Mean Placebo-adjusted Change of PR from Baseline at Various Edaravone Concentration Levels and 2-sided 90% Confidence Bounds (msec) at Various Edaravone Concentration Levels and 2-sided 90% Confidence Bounds (msec) at Various Edaravone Concentration Levels and 2-sided 90% Confidence Bounds (msec)

Table 11: Edaravone QTcF Regression Analysis: Regression Statistics

| O.F. | AIC | | | |
|------|-------|--------|-----------|-------|
| | Model | Linear | Quadratic | Cubic |

Repeat as:

Table 12: Edaravone HR Regression Analysis: Regression Statistics Table 13: Edaravone PR Regression Analysis: Regression Statistics Table 14: Edaravone QRS Regression Analysis: Regression Statistics

Table 15: LS Mean Changes from Baseline in QTcF for Edaravone and Placebo and LS Mean Placebo-subtracted Changes from Baseline in QTcF and two-sided 90% Upper Confidence Bounds (msec)

| | | Edara | Edaravone | Combine | Combined Placebo | Edara | Edaravone - Placebo |
|---|---|---|---|---|---|---|---|
| Treatment | Timepoint (hrs postdose) | z | LS Mean | Z | LS Mean | ΔΔQΤcF | Two-sided 90%<br>CI Upper Bound |
| | 0.25 | | | | | | |
| | 0.5 | | | | | | |
| | П | | | | | - | |
| | 1.5 | | | | | | |
| Edaravone | 2 | | | | | | * |
| 300 mg | 4 | | | | | | |
| with | 9 | | | | | | |
| xanthan PO | 8 | | | | | | |
| | 12 | | - | | | | |
| | 24 | | | | | | |
| | 36 | | | | | | |
| | 48 | | | | | | |
| | 0.25 | | | | | | |
| | 0.5 | | | | | | |
| | | - | | | | | |
| Edaravone | 1.5 | - | | | • | | |
| 300 mg | 2 | 5 | | | | | |
| withiout | 4 | | | | | | |
| | 9 | | - | | | | |
| | 8 | | | | | | |
| | 12 | | | | | | |


| | | | | Ţ | | | | | | | | | | | . [ | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Edaravone - Placebo | Two-sided 90%<br>CI Upper Bound | | | | | | | į | | | | | | | | |
| Edara | AAQTCF | | | - | | | | | | | | | | | | |
| Combined Placebo | LS Mean | · | | | | | | | | | | | | | | |
| Combine | Z | | | | | | | | | | | | | | | |
| vone | LS Mean | | | | | | | | | | | - | | | | |
| Edaravone | Z | | | | | | | | | | | | | | | |
| | Timepoint (hrs postdose) | 24 | 36 | 48 | 0.25 | 0.5 | H | 1.5 | 2 | 4 | 9 | 8 | 12 | 24 | 36 | 48 |
| | Treatment | | | | | | | • | • | Edaravone | 30 mg | | | | | |

Repeat as:

Table 16: LS Mean Changes from Baseline for HR for Edaravone and Placebo and LS Mean Placebo-subtracted Changes from Baseline in QTcF and 2-sided 90% Upper Confidence Bounds (msec)

Table 17: LS Mean Changes from Baseline for PR for Edaravone and Placebo and LS Mean Placebo-subtracted Changes from Baseline in QTcF and 2-sided 90% Upper Confidence Bounds (msec)

Table 18: LS Mean Changes from Baseline for QRS for Edaravone and Placebo and LS Mean Placebo-subtracted Changes from Baseline in QTcF and 2-sided 90% Upper Confidence Bounds (msec)


Table 19: Number (%) of Subjects with a QTcF Interval >450 msec

| | | | | 3 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Comb | Combined Placebo | oqeo | Edara<br>with | Edaravone 300 mg<br>with xanthan PO | 00 mg<br>n Po | Edara | Edaravone 300 mg<br>without xanthan<br>PO | o mg<br>than | Edara<br>so | Edaravone30 mg<br>solution PO | o mg |
| Timepoint (hrs postdose) | z | ב | % | Z | n | % | z | ב | % | z | u | % |
| Baseline | | | | | | | | | | | | |
| 0.25 | | | | | | | | | | | | |
| 0.5 | | | | | | | | ÷ | | | | |
| 1 | | | | | | | | | | | | |
| 1.5 | | | | | | | | | | | | |
| 2 | | | | | | | | | | | | |
| 4 | | | | | | | | | | | | |
| 9 | | | | | | | | | | | | |
| 8 | | | | | | | | | | | | |
| 12 | | | | | | | | | | | | |
| 24 | | | | | | | | | - | | | |
| 36 | | | | | | ļ | | | | | | |
| 48 | | | | | : | | | | | | | |
| Overall | | | | | | | | | | | | } |

# MITSUBISHI TANABE PHARMA CORPORATION CONFIDENTIAL

Repeat Table 15 as:

Table 20: Number (%) of Subjects with a QTcF Interval >480

Table 21: Number (%) of Subjects with a QTcF Interval >500 msec

Table 22: Number (%) of Subjects with a QTcF Interval Change from Baseline in QTcF >30 msec

Table 24: Number (%) of Subjects with HR <40 bpm after a decrease of HR ≥20 bpm from Baseline Table 23: Number (%) of Subjects with a QTcF Interval Change from Baseline in QTcF >60 msec

Table 25: Number (%) of Subjects with HR >110 bpm after an increase of HR >20 bpm from Baseline

Table 27: Number (%) of Subjects with PR interval of >220 msec after an increase of PR interval ≥25% from Baseline Table 26: Number (%) of Subjects with PR interval of <100 msec after a decrease of PR interval ≥25% from Baseline

Table 28: Number (%) of Subjects with QRS duration >120 msec after an increase of QRS duration ≥25% from Baseline


Table 29: Subjects with an ECG Diagnostic Finding Not Present at Baseline Tracings

| | , | | 0 | | ) | | | | | , | | | г |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Over All Timepoint | Combi | Combined Placebo | oqeou | Edara\<br>with | Edaravone 300 mg<br>with xanthan PO | 00 mg<br>n PO | Edarav | Edaravone 300 mg<br>without xanthan<br>PO | 0 mg<br>than | Edara<br>So | Edaravone30 mg<br>solution PO | 0 mg | - |
| Finding | z | u | % | Z | u | % | z | ב | % | z | u | % | |
| Finding 1 | | | | | | | | | | | | | - |
| Finding 2 | | | | | | | | | | | | | - |
| etc. | | | | | | | | | | | | | |

Figure 2: Arithmetic Mean QTcF (msec)



Figure 3: Arithmetic Mean HR (bpm) Figure 4: Arithmetic Mean PR (msec) Figure 5: Arithmetic Mean QRS (msec)

Repeat as:

Figure 6: Arithmetic Mean Change from Baseline in QTcF



Figure 7: Arithmetic Mean Change from Baseline in HR (bpm) Figure 8: Arithmetic Mean Change from Baseline in PR (msec) Figure 9: Arithmetic Mean Change from Baseline in QRS (msec)

Repeat as:

Figure 10: Edaravone QTcF-Concentration Regression Analysis: Change of QTcF from Baseline versus Edaravone Concentration, Combined Doses: Slope (if linear) and 2-sided 90% Confidence Bounds of the Slope (msec)



Repeat Figure 9 as:

Figure 13: Edaravone QRS-Concentration Regression Analysis: Change of QTcF from Baseline versus Edaravone Figure 11: Edaravone HR-Concentration Regression Analysis: Change of QTcF from Baseline versus Edaravone Figure 12: Edaravone PR-Concentration Regression Analysis: Change of QTcF from Baseline versus Edaravone Concentration, Combined Doses: Slope (if linear) and 2-sided 90% Confidence Bounds of the Slope (msec) Concentration, Combined Doses: Slope (if linear) and 2-sided 90% Confidence Bounds of the Slope (msec) Concentration, Combined Doses: Slope (if linear) and 2-sided 90% Confidence Bounds of the Slope (msec)

Figure 14: Edaravone QTcF-Concentration Regression Analysis: From Slope and 2-sided 90% Confidence Bounds of the Slope (if linear), Combined Doses: Estimated Mean Placebo-adjusted Change of QTcF from Baseline at Geometric Mean



X axis will be 3 points only, labelled as: "Geometric Mean Cmax (ng/mL)" - "Edaravone 300 mg with Xanthan PO" "Edaravone 300 mg without Xanthan PO" "Edaravone 30 mg solution PO"

Figure 15: Edaravone HR-Concentration Regression Analysis: From Slope (if linear) and 2-sided 90% Confidence Bounds of the Slope, Combined Doses: Estimated Mean Placebo-adjusted Change of QTcF from Baseline at Geometric Mean Cmax Edaravone Concentration Levels and 2-sided 90% Confidence Bounds (msec)

Figure 16: Edaravone PR-Concentration Regression Analysis: From Slope (if linear) and 2-sided 90% Confidence Bounds of the Slope, Combined Doses: Estimated Mean Placebo-adjusted Change of QTcF from Baseline at Geometric Mean Cmax Edaravone Concentration Levels and 2-sided 90% Confidence Bounds (msec)

Figure 17: Edaravone QRS-Concentration Regression Analysis: From Slope (if linear) and 2-sided 90% Confidence Bounds of the Slope, Combined Doses: Estimated Mean Placebo-adjusted Change of QTcF from Baseline at Geometric Mean Cmax Edaravone Concentration Levels and 2-sided 90% Confidence Bounds (msec)

Figure 18: Change of HR from Baseline versus Edaravone Concentration and 2-sided 90% Confidence Bounds of the Slope (msec)



Y axis will be Change of HR (bpm)

Figure 19: QTcF vs. RR and 2-sided 90% Confidence Bounds of the Slope (msec)



X-axis will be RR (bpm), Y axis will be QTcF (msec)

Figure 20: Hysteresis Analysis: Highest Edaravone Dose Group: LS Mean Placebo-adjusted Change from Baseline (ΔΔQTcF)



Figure 21: Paired AQTc and Concentration with Loess Smooth Line and 95% Confidence Intervals and Linear Regression



Repeat as:

Figure 24: Paired AQRS and Concentration with Loess Smooth Line and 95% Confidence Intervals and Linear Regression Figure 22: Paired A HR and Concentration with Loess Smooth Line and 95% Confidence Intervals and Linear Regression Figure 23: Paired APR and Concentration with Loess Smooth Line and 95% Confidence Intervals and Linear Regression

MITSUBISHI TANABE PHARMA CORPORATION CONFIDENTIAL

Figure 25: Edaravone QTcF-Concentration Regression Analysis: Model Predicted vs Observed AQTcF Figure 28: Edaravone QRS-Concentration Regression Analysis: Model Predicted vs Observed AQRS Figure 26: Edaravone HR-Concentration Regression Analysis: Model Predicted vs Observed AQHR Figure 27: Edaravone PR-Concentration Regression Analysis: Model Predicted vs Observed APR

Figure 31: Edaravone PR-Concentration Regression Analysis: Quantile-Quantile Plot of Residuals Concentration Figure 29: Edaravone QTcF-Concentration Regression Analysis: Quantile-Quantile Plot of Residuals Figure 32: Edaravone QRS-Concentration Regression Analysis: Quantile-Quantile Plot of Residuals Figure 30: Edaravone HR-Concentration Regression Analysis: Quantile-Quantile Plot of Residuals

Figure 33: Edaravone QTcF-Concentration Regression Analysis: Concentration vs Residuals Figure 36: Edaravone QRS-Concentration Regression Analysis: Concentration vs Residuals Figure 34: Edaravone HR-Concentration Regression Analysis: Concentration vs Residuals Figure 35: Edaravone PR-Concentration Regression Analysis: Concentration vs Residuals

Figure 40: Edaravone QRS Regression Analysis: Baseline QRS vs Residuals Residuals Figure 37: Edaravone QTcF Regression Analysis: Baseline QTcF vs Residuals Figure 38: Edaravone HR Regression Analysis: Baseline HR vs Residuals Figure 39: Edaravone PR Regression Analysis: Baseline PR vs Residuals

Figure 41: Edaravone QTcF Regression Analysis: Active Treatment vs Residuals Figure 42: Edaravone HR Regression Analysis: Active Treatment vs Residuals Figure 43: Edaravone PR Regression Analysis: Active Treatment vs Residuals Figure 44: Edaravone QRS Regression Analysis: Active Treatment vs Residuals

Figure 45: LS Mean Placebo-adjusted Change from Baseline in QTcF and 1-sided Upper 95% Confidence Bounds (msec)



# Repeat as:

Figure 48: LS Mean Placebo-adjusted Change from Baseline in QRS and 2-sided 90% CIs Confidence Bounds (msec) Figure 47: LS Mean Placebo-adjusted Change from Baseline in PR and 2-sided 90% CIs Confidence Bounds (msec) Figure 46: LS Mean Placebo-adjusted Change from Baseline in HR and 2-sided 90% CIs Confidence Bounds (bpm)

Appendix 1: Listing of Individual Subject ECG Data

| | , |
|----------------|---------|
| QTcF | (msec) |
| QT | (msec) |
| QRS | (msec) |
| PR | (msec) |
| RR | (msec) |
| 光 | (mdq) |
| Time | ) |
| Dose | Group |
| Cohort | |
| Subject Cohort | Janjeer |

Note: intervals are means of all Baseline ECGs or of triplicate ECGs at postdose timepoints


Appendix 2: Listing of Individual Subject Change of ECG Intervals ( $\Delta$ ) and Edaravone Concentration

| Cohort Group Time (bpm) (msec) (msec) | | | Dose | | H | PR | ORS | OTCF | Concentration |
|---|---|---|---|---|---|---|---|---|---|
| | Subject | Cohort | Group | Time | (pbm) | (msec) | (msec) | (msec) | (ng/mL) |
| | | | | | | | - | : | |
| | | | | | | ٠ | | | |

Note: interval changes are means of triplicate ECGs. Concentration values for Placebo will be null. Concentrations below level of quantitation or not detectable for edaravone will be set to 0.

Appendix 3: Listing of Abnormal ECG Morphologies

| Emergent<br>from<br>Baseline<br>(Y/N) |
|---------------------------------------|
| Finding |
| Time |
| t Group Time |
| Cohort |
| Subject Cohort |

Note: findings are those on any of the Baseline ECGs or on any of triplicate ECGs at postdose timepoints